CLINICAL TRIAL: NCT00412984
Title: A Phase 3, Active (Warfarin) Controlled, Randomized, Double-Blind, Parallel Arm Study to Evaluate Efficacy and Safety of Apixaban in Preventing Stroke and Systemic Embolism in Subjects With Nonvalvular Atrial Fibrillation
Brief Title: Apixaban for the Prevention of Stroke in Subjects With Atrial Fibrillation
Acronym: ARISTOTLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV185-030
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2013-04-29 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-05

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Warfarin; apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: warfarin
- 2 (Experimental)
  Interventions: Drug: apixaban

INTERVENTIONS:
Drug: warfarin — Oral tablets, 2.0 mg, adjusted to an INR of 2.5 (range 2.0 to 3.0)
  Other Names: Coumadin; BMS-565793
  Arms: 1
Drug: apixaban — Oral tablets, 5.0 mg or 2.5 mg, twice daily
  Other Names: BMS-562247
  Arms: 2

SUMMARY:
The trial seeks to determine if apixaban, an investigational anticoagulant (blood-thinner) is as effective as standard therapy (warfarin) in preventing stroke and systemic embolism in subjects with atrial fibrillation and risk factors for stroke.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 yrs with atrial fibrillation (AF) and one or more of the following risk factors for stroke:
* Age ≥ 75, previous stroke
* transient ischemic attack (TIA) or Systemic Embolism (SE)
* Symptomatic congestive heart failure or left ventricular dysfunction with left ventricular ejection fraction (LVEF) ≤ 40%
* Diabetes mellitus or hypertension requiring pharmacological treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20976 (Actual)
Dates: Start 2006-12-31 (Actual); Primary Completion 2011-05-25 (Actual); Study Completion 2011-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (829):
- United States (271):
  - Cardiovascular Associates, Pc, Birmingham, Alabama
  - Alabama Internal Medicine Pc, Birmingham, Alabama
  - Birmingham Heart Clinic P.C., Birmingham, Alabama
  - Heart Center, Inc., Huntsville, Alabama
  - Mobile Heart Specialists, Pc, Mobile, Alabama
  - Clara V. Massey, Md, Mobile, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Internal Medicine Physicians Associates, P.C., Phoenix, Arizona
  - Southwest Heart, Tucson, Arizona
  - Southern Arizona Va Health Care System, Tucson, Arizona
  - Pima Research Foundation, Tucson, Arizona
  - Dr. Rajesh Shroff, Hot Springs, Arkansas
  - Mary K. Richards, Md Pa, Little Rock, Arkansas
  - Advanced Clinical Reserach Institute, Anaheim, California
  - Act/Cardiovascular Research Institute, Beverly Hills, California
  - Capitol Interventional Cardiology, Carmichael, California
  - Escondido Cardiology Associates, Inc., Escondido, California
  - William D. Bowden, D.O., Healdsburg, California
  - La Mesa Cardiac Center, A Medical Group, La Mesa, California
  - Va Greater Los Angeles Healthcare System, Los Angeles, California
  - Coastal Cardiology, Mission Viejo, California
  - Kenneth W. Carr Md, Oceanside, California
  - Desert Med Grp Inc, Dba Desert Oasis Healthcare Med Group, Palm Springs, California
  - Desert Cardiology Consultants Medical Group, Inc, Rancho Mirage, California
  - Regional Cardiolody Associates, Sacramento, California
  - Northern California Research, Sacramento, California
  - Sacramento Heart And Vascular Medical Associates, Sacramento, California
  - Arrhythmia Consultants Of The Central Coast Medical Group, Santa Barbara, California
  - Northern California Medical Associates, Santa Rosa, California
  - Progressive Clinical Research, Vista, California
  - Cardivasclular Consultants Medical Group, Walnut Creek, California
  - Shiva Heart Center Medical Group, Wildomar, California
  - Electrophysiology Associates, Pc, Colorado Springs, Colorado
  - Aurora Denver Cardiology Associates, P.C., Denver, Colorado
  - Denver Va Medical Center, Denver, Colorado
  - New West Physicians Clinical Research, Golden, Colorado
  - South Denver Cardiology Associates Pc, Littleton, Colorado
  - Connecticut Clinical Research, Llc, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Cardiology Associates Of New Haven,Pc, Guilford, Connecticut
  - The William W. Backus Hospital, Norwich, Connecticut
  - William W Backus Hospital, Norwich, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Chase Medical Research, Llc, Waterbury, Connecticut
  - Alfieri Cardiology, Newark, Delaware
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Washington Va Medical Center, Washington D.C., District of Columbia
  - Medical Specialist Of The Palm Beach, Atlantis, Florida
  - Miami International Cardiology Consultants, Aventura, Florida
  - David Charles Mishkel, Md, Pa, Boca Raton, Florida
  - The Heart & Vascular Institute Of Florida, Clearwater, Florida
  - The Heart And Vascular Institute Of Florida, Clearwater, Florida
  - Cardiovascular Specialist Of South Florida, Davie, Florida
  - Daytona Heart Group, Daytona Beach, Florida
  - Cardiology Associates Of Fort Lauderdale, P.A., Fort Lauderdale, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Florida Heart Associates, Fort Myers, Florida
  - Florida Research Network, Llc, Gainesville, Florida
  - Healthworx, Hollywood, Florida
  - Luis Tami, Md, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - St. Vincent'S Ambulatory Care, Inc, Jacksonville, Florida
  - Jacksonville Heart Center, Pa, Jacksonville, Florida
  - Jacksonville Cardiovascular Center, Jacksonville, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - St. Luke'S Cardiology, Jacksonville, Florida
  - Jacksonville Heart Center, P.A., Jacksonville Beach, Florida
  - Cvms Research Institute, Llc, Jupiter, Florida
  - Ricardo Bedoya, M.D., Jupiter, Florida
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Miami International Cardiology Consultants, Miami, Florida
  - Physicians Regional Medical Group, Naples, Florida
  - Florida Heart Group, Orlando, Florida
  - Alpha Medical Research, Oviedo, Florida
  - Cardiology Consultants, Pensacola, Florida
  - Niranjan Seshadri, Md, Sarasota, Florida
  - Heart & Vascular Center Research, Inc., Sarasota, Florida
  - The Heart And Vascular Institute Of Florida, St. Petersburg, Florida
  - Research, Inc., Vero Beach, Florida
  - Cardiovascular Specialits, Pc, Atlanta, Georgia
  - Augusta Cardiology Clinic, P.C., Augusta, Georgia
  - Columbus Cardiology Associates Pc, Columbus, Georgia
  - Columbus Cardiology Associates,Pc, Columbus, Georgia
  - Georgia Heart Specialists, L.L.C., Covington, Georgia
  - Atlanta Institute For Medical Research, Inc, Decatur, Georgia
  - Northeast Georgia Heart Center, Pc, Gainesville, Georgia
  - Wellstar Cardiovascular Medicine, Pc, Marietta, Georgia
  - Fox Valley Clinical Research Center, Llc, Aurora, Illinois
  - Nmff, Chicago, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois Heart & Lung Research Center, Sc, Normal, Illinois
  - Cpt. James A Lovell Federal Health Care Center, North Chicago, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Premier Healthcare, Llc, Bloomington, Indiana
  - Elkhart Clinic, Llc, Elkhart, Indiana
  - Lutheran Medical Group, Llc, Fort Wayne, Indiana
  - Fort Wayne Cardiology, Fort Wayne, Indiana
  - St Francis Medical Group - Indiana Heart Physicians, Indianapolis, Indiana
  - The Care Group, Llc., Indianapolis, Indiana
  - The Care Group, Llc, Indianapolis, Indiana
  - Dali, Sammi, Michigan City, Indiana
  - Cardiology Associates, Inc., South Bend, Indiana
  - Mcfarland Clinic Pc, Ames, Iowa
  - Midwest Cardiology Associates , P.C., Overland Park, Kansas
  - Central Cardiology Assoc., Elizabethtown, Kentucky
  - New Lexington Clinic, P.S.C., Lexington, Kentucky
  - Va Medical Center, Louisville, Kentucky
  - Norton Cardiovascular Associates, Louisville, Kentucky
  - Owensboro Heart & Vascular, Owensboro, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Cardiovascular Institute Of The South, Houma, Louisiana
  - Smith, Patel & Amkieh, Llc, Lacombe, Louisiana
  - Imperial Calcasieu Medical Group, Llp, Lake Charles, Louisiana
  - Cardiology Center, Llc, Marrero, Louisiana
  - Cardiology Associates, Shreveport, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Medical Research Inst, Inc, Slidell, Louisiana
  - Medical Research Institute, Inc, Slidell, Louisiana
  - Ventura Cardio. Cond. Med. Group, Inc., Ventura, Louisiana
  - Central Maine Heart & Vascular Institute, Lewiston, Maine
  - Midatlantic Cardiovascular Associates, P.A., Baltimore, Maryland
  - Midatlantic Cardiovascular Associates, Pa, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Franklin Square Hospital, Baltimore, Maryland
  - Midatlantic Cardiovascular Associates, Pa, Bel Air, Maryland
  - Cardiovascular Specialists Of Central Maryland, P.A., Columbia, Maryland
  - Clinical Associates Research, Reisterstown, Maryland
  - Midatlantic Cardiovascular Associates, Pa, Westminster, Maryland
  - Burlington Medical Associates, Billerica, Massachusetts
  - Caritas St. Elizabeth'S Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Neccr Internal Medicine & Cardiology Associates,Llc, Fall River, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Charles River Medical Associates, Natick, Massachusetts
  - Great Lakes Heart Center Of Alpena, Alpena, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Thoracic And Cardiovascular Healthcare Foundation, Lansing, Michigan
  - Advanced Cardiovascular Health Specialists, Pc, Livonia, Michigan
  - Michigan Heart And Vascular Specialists, Petoskey, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Heart, P.C., Ypsilanti, Michigan
  - Minneapolis Va Medical Center, Minneapolis, Minnesota
  - University Of Minnesota, Minneapolis, Minnesota
  - North Memorial Health Care, Robbinsdale, Minnesota
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Tupelo Neurology Clinic, Pa, Tupelo, Mississippi
  - University Of Missouri, Columbia, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke'S Lipid And Diabetes Research Center, Kansas City, Missouri
  - Internal Medical Associates of Grand Island, P.C, Grand Island, Nebraska
  - Internal Medical Associates Of Grand Island, P.C, Grand Island, Nebraska
  - Nebraska Heart Institute, Hastings, Nebraska
  - Va Southern Nevada Healthcare System, Las Vegas, Nevada
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Cardiovascular Associates Of The Delware Valley, P.A., Elmer, New Jersey
  - Cardiovascular Associates Of The Delaware Valley, P.A., Haddon Heights, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Cardio Assoc Of Del Val, P.A., Sewell, New Jersey
  - Central New Jersey Cardiology, South Plainfield, New Jersey
  - Abq Health Partners, Llc, Albuquerque, New Mexico
  - University Of New Mexico/University Hospital, Albuquerque, New Mexico
  - Albany Assoc. In Cardiology, Albany, New York
  - Albany Associates In Cardiology, Albany, New York
  - Cardiology Associates, Pc, Binghamton, New York
  - Buffalo Heart Group, Llp, Buffalo, New York
  - Bruce L. Platt Md, Pc, Buffalo, New York
  - Bruce L. Platt, Md, Buffalo, New York
  - Heart Care Center, P.C., East Syracuse, New York
  - Huntington Hospital, Huntington, New York
  - Sjh Cardiology Associates, Liverpool, New York
  - Long Island Heart Associates, Mineola, New York
  - Saratoga Cardiology Associates, Pc, Saratoga Springs, New York
  - Office Of Dr. Kozinn, Williamsville, New York
  - Suburban Cardiology, Williamsville, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Kernodle Clinic, Inc., Burlington, North Carolina
  - Carolina Cardiology Associates, Pa, High Point, North Carolina
  - Pinehurst Medical Center, Inc, Pinehurst, North Carolina
  - Lillestol Research Llc, Fargo, North Dakota
  - Akron Cardiology Consultants, Akron, Ohio
  - Christopher M. Johnson, D.O., Bucyrus, Ohio
  - Community Health Care, Inc., Canal Fulton, Ohio
  - Cardiology Associates, Canton, Ohio
  - The Carl & Edyth Lindner Center For R&E At The Christ Hosp, Cincinnati, Ohio
  - Toledo Cardiology Consultants, Toledo, Ohio
  - Family Practice Center Of Wadsworth, Inc., Wadsworth, Ohio
  - Jack C. Va Medical Center, Muskogee, Oklahoma
  - Cor Clinical Research, Llc, Oklahoma City, Oklahoma
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Plaza Medical Group, Pc, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Physicians, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Eminence Research, Llc, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Consultants, Llc, Tulsa, Oklahoma
  - St. Charles Health System, Inc., Bend, Oregon
  - St. Charles Health System, Inc, Bend, Oregon
  - Oregon Medical Group - Clinical Research, Eugene, Oregon
  - Hillsboro Cardiology Pc, Hillsboro, Oregon
  - Rogue Valley Physicians - Clinical Research Group, Medford, Oregon
  - Abington Medical Specialists, Abington, Pennsylvania
  - Blair Medical Associates, Inc., Altoona, Pennsylvania
  - Heritage Cardiology Assoc., Camp Hill, Pennsylvania
  - Central Bucks Cardiology, Doylestown, Pennsylvania
  - Internal Medicine And Lipid Mgmt., Erie, Pennsylvania
  - Kandra, Fierer, Kuskin Associates, Harrisburg, Pennsylvania
  - Pivotal Clinical Research, Llc, Hatfield, Pennsylvania
  - Lycoming Internal Medicine Inc., Jersey Shore, Pennsylvania
  - Guthrie Clinic Ltd., Sayre, Pennsylvania
  - Guthrie Medical Group, P.C., Sayre, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - West Chester Cardiology, Pc, West Chester, Pennsylvania
  - Cardiology Consultants Of Philadelphia, Yardley, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Southeastern Research Associates, Inc, Anderson, South Carolina
  - Lowcountry Medical Group, Llc, Beaufort, South Carolina
  - Lowcountry Medical Group, Beaufort, South Carolina
  - Medical University Of South Carolina, Charleston, South Carolina
  - Columbia Heart Clinic, Columbia, South Carolina
  - Upstate Cardiology, Greenville, South Carolina
  - Internal Medicine Of Greer, Greer, South Carolina
  - Palmetto Nephrology Pa, Orangeburg, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Avera Medical Associates Clinic, Pierre, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Knoxville Heart Group, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Tennessee Center For Clinical Trials, Tullahoma, Tennessee
  - Amarillo Heart Clinical Research Institute Inc., Amarillo, Texas
  - Corsicana Medical Research, Pllc, Corsicana, Texas
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - Heartplace, Dallas, Texas
  - Heart Center Of North Texas, Fort Worth, Texas
  - Center For Atrial Fibrillation, Houston, Texas
  - The Methodist Hospital Neurology Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - Northwest Houston Cardiology, Pa, Houston, Texas
  - Francisco R. Maislos, Houston, Texas
  - Woodlands North Houston Heart Center, Houston, Texas
  - Regional Medical Center And Diagnostic Clinics, Humble, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Dcol Center For Clinical Research, Longview, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Legacy Heart Center, Plano, Texas
  - North Texas Medical Research, Plano, Texas
  - Bhs Specialty Network, Inc, San Antonio, Texas
  - Covenant Clinical Research, Pa, San Antonio, Texas
  - Star Clinical Trails, San Antonio, Texas
  - Edward Balli, Md, Pa, Seguin, Texas
  - Northwest Heart Center, Tomball, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - The Univ. Of Texas Health Science Ctr. At Tyler, Tyler, Texas
  - University Of Texas Health Science Center At Tyler, Tyler, Texas
  - Utah Cardiology P.C, Layton, Utah
  - Sentara York Clinical Research, Norfolk, Virginia
  - Medical Research Initiatives, Richmond, Virginia
  - Roanoke Heart Institute, Plc, Roanoke, Virginia
  - Cardiovascular Associates, Virginia Beach, Virginia
  - Daniel W. Gottlieb, Md, Ps, Burien, Washington
  - Daniel William Gottlieb, Md, Burien, Washington
  - Rockwood Clinic Research Cent., Spokane, Washington
  - Walla Walla Clinic, Walla Walla, Washington
  - Lynn N. Smith, Md, Lewisburg, West Virginia
  - Cardiology Associates Of Green Bay Ltd-Bellin Hospital, Green Bay, Wisconsin
  - St. Mary'S Hospital, Madison, Wisconsin
  - St.Mary'S Hospital, Madison, Wisconsin
  - Aurora Health Care, Milwaukee, Wisconsin
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
  - Cardiology Assc. Of Waukesha, Waukesha, Wisconsin
- Argentina (27):
  - Local Institution, Adrogué, Buenos Aires
  - Local Institution, Bahía Blanca, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution, Ciudad Autonoma de, Buenos Aires
  - Local Institution, Ciudad Autonoma, Buenos Aires
  - Local Institution, Coronel Suárez, Buenos Aires
  - Local Institution, Haedo, Buenos Aires
  - Local Institution, Junín, Buenos Aires
  - Local Institution, La Plata, Buenos Aires
  - Local Institution, Mar del Plata, Buenos Aires
  - Local Institution, Merlo, Buenos Aires
  - Local Institution, Olivos, Buenos Aires
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Ramos Mejía, Buenos Aires
  - Local Institution, San Justo, Buenos Aires
  - Local Institution, San Martín, Buenos Aires
  - Local Institution, San Nicolás de los Arroyos, Buenos Aires
  - Local Institution, Zárate, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Cipolletti, Río Negro Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miquel de Tucuman, Tucumán Province
  - Local Institution, Buenos Aires
  - Local Institution, Córdoba
  - Local Institution, Salta
  - Local Institution, San Miguel de Tucumán
  - Local Institution, Santa Fe
- Australia (21):
  - Local Institution, Coffs Harbour, New South Wales
  - Local Institution, Concord, New South Wales
  - Local Institution, Gosford, New South Wales
  - Local Institution, Kogarah, New South Wales
  - Local Institution, Miranda, New South Wales
  - Local Institution, Auchenflower, Queensland
  - Local Institution, Brisbane, Queensland
  - Local Institution, Caboolture, Queensland
  - Local Institution, Herston, Queensland
  - Local Institution, Kippa-Ring, Queensland
  - Local Institution, Nambour, Queensland
  - Local Institution, Sherwood, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Ashford, South Australia
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Woodville, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Dandenong, Victoria
  - Local Institution, Geelong, Victoria
  - Local Institution, Fremantle, Western Australia
  - Local Institution, Joondalup, Western Australia
- Austria (3):
  - Local Institution, Graz
  - Local Institution, Oberpullendorf
  - Local Institution, Vienna
- Belgium (18):
  - Local Institution, Aalst
  - Local Institution, Antwerp
  - Local Institution, Arlon
  - Local Institution, Bruges
  - Local Institution, Brussels
  - Local Institution, Dillingen
  - Local Institution, Genk
  - Local Institution, Ghent
  - Local Institution, Gilly
  - Local Institution, Hasselt
  - Local Institution, Huy
  - Local Institution, Kortrijk
  - Local Institution, Menen
  - Local Institution, Mol
  - Local Institution, Montegnée
  - Local Institution, Verviers
  - Local Institution, Woluwe-Saint-Lambert
  - Local Institution, Yvoir
- Brazil (22):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Belo Horzonte, Minas Gerais
  - Local Institution, Juiz de Fora, Minas Gerais
  - Local Institution, Uberaba, Minas Gerais
  - Local Institution, Uberlândia, Minas Gerais
  - Local Institution, Campina Grande do Sul, Paraná
  - Local Institution, Curitiba, Paraná
  - Local Institution, Londrina, Paraná
  - Local Institution, Belém, Pará
  - Local Institution, Natal, Rio Grande do Norte
  - Local Institution, Porte Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Blumenau, Santa Catarina
  - Local Institution, São José, Santa Catarina
  - Local Institution, Botucatu, São Paulo
  - Local Institution, Campinas, São Paulo
  - Local Institution, Marília, São Paulo
  - Local Institution, San Jose Do Rio Preto, São Paulo
  - Local Institution, Santo André, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (39):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Burnaby, British Columbia
  - Local Institution, Nanaimo, British Columbia
  - Local Institution, New Westminster, British Columbia
  - Local Institution, North Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Brampton, Ontario
  - Local Institution, Burlington, Ontario
  - Local Institution, Cambridge, Ontario
  - Local Institution, Greater Sudbury, Ontario
  - Local Institution, Hamilton, Ontario
  - Local Institution, London, Ontario
  - Local Institution, Mississauga, Ontario
  - Local Institution, Newmarket, Ontario
  - Local Institution, Niagara Falls, Ontario
  - Local Institution, North Bay, Ontario
  - Local Institution, Oshawa, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Scarborough Village, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Weston, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Drummondville, Quebec
  - Local Institution, Greenfield Park, Quebec
  - Local Institution, Lachine, Quebec
  - Local Institution, Lévis, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Pointe-Claire, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Saint-Lambert, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Chile (5):
  - Local Institution, Osorno, Los Lagos Region
  - Local Institution, Temuco, Región de la Araucanía
  - Local Institution, Temuco, Región de Valparaíso
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Santiago, Santiago Metropolitan
- China (18):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Lanzhou, Gansu
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Shijiazhuang, Hebei
  - Local Institution, Daqing, Heilongjiang
  - Local Institution, Haerbin, Heilongjiang
  - Local Institution, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Hangzhou, Jiangsu
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Dalian, Liaoning
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Jinan, Shandong
  - Local Institution, Qingdao, Shandong
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Chongqing, Sichuan
  - Local Institution, Hangzhou, Zhejiang
- Colombia (5):
  - Local Institution, Medellín, Antioquia
  - Local Institution, Barranquilla
  - Local Institution, Bogotá
  - Local Institution, Cali
  - Local Institution, Medellín
- Czechia (11):
  - Local Institution, Boskovice
  - Local Institution, Brno
  - Local Institution, Brno-Malomerice
  - Local Institution, Ivančice
  - Local Institution, Kladno
  - Local Institution, Litomyšl
  - Local Institution, Městec Králové
  - Local Institution, Ostrava
  - Local Institution, Prague
  - Local Institution, Příbram
  - Local Institution, Ústí nad Orlicí
- Denmark (17):
  - Local Institution, Arhus C
  - Local Institution, Copenhagen
  - Local Institution, Esbjerg
  - Local Institution, Frederiksberg
  - Local Institution, Frederikssund
  - Local Institution, Gentofte Municipality
  - Local Institution, Haderslev
  - Local Institution, Hellerup
  - Local Institution, Herlev
  - Local Institution, Herning
  - Local Institution, Hillerød
  - Local Institution, Hvidovre
  - Local Institution, Kolding
  - Local Institution, Odense
  - Local Institution, Silkeborg
  - Local Institution, Slagelse
  - Local Institution, Svendborg
- Finland (7):
  - Local Institution, Helsinki
  - Local Institution, Hus
  - Local Institution, Jyväskylä
  - Local Institution, Kemi
  - Local Institution, Oulu
  - Local Institution, Pori
  - Local Institution, Tampere
- France (7):
  - Local Institution, Amiens
  - Local Institution, Bordeaux
  - Local Institution, Brest
  - Local Institution, Grenoble
  - Local Institution, La Seyne-sur-Mer
  - Local Institution, Paris
  - Local Institution, Six-Fours-les-Plages
- Germany (34):
  - Local Institution, Aachen
  - Local Institution, Bad Krozingen
  - Local Institution, Bad Neustadt/ Salle
  - Local Institution, Bad Oeynhausen
  - Local Institution, Berlin
  - Local Institution, Betzdorf
  - Local Institution, Bochum
  - Local Institution, Bonn
  - Local Institution, Coburg
  - Local Institution, Dillingen
  - Local Institution, Dresden
  - Local Institution, Duisburg
  - Local Institution, Essen
  - Local Institution, Frankfurt am Main
  - Local Institution, Göttingen
  - Local Institution, Halle
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Kassel
  - Local Institution, Köpenick
  - Local Institution, Lahr
  - Local Institution, Ludwigshafen
  - Local Institution, Mannheim
  - Local Institution, Marburg
  - Local Institution, München
  - Local Institution, Osnabrück
  - Local Institution, Regensburg
  - Local Institution, Riesa
  - Local Institution, Rostiock
  - Local Institution, Trier
  - Local Institution, Waren
  - Local Institution, Witten
  - Local Institution, Wolmirstedt
  - Local Institution, Worms
- Hong Kong (2):
  - Local Institution, Hong Kong
  - Local Institution, Shatin
- Hungary (14):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Dunaújváros
  - Local Institution, Győr
  - Local Institution, Gyula
  - Local Institution, Hódmezővásárhely
  - Local Institution, Komárom
  - Local Institution, Mosonmagyaróvár
  - Local Institution, Orosháza
  - Local Institution, Pécs
  - Local Institution, Siófok
  - Local Institution, Sopron
  - Local Institution, Szentes
  - Local Institution, Zalaegerszeg
- India (29):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Visakhapatnam, Andhra Pradesh
  - Local Institution, Visakhapatnam, Andhrapradesh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Vadodara, Gujarat
  - Local Institution, Bangalore, Karnataka
  - Local Institution, Mysore, Karnataka
  - Local Institution, Calicut, Kerala
  - Local Institution, Pune, Maharashta
  - Local Institution, Nagpur, Maharashtra
  - Local Institution, Pune, Maharashtra
  - Local Institution, Jalandhar, Punjab
  - Local Institution, Bikaner, Rajasthan
  - Local Institution, Lucknow, Uttar Pradesh
  - Local Institution, Ahmedabad
  - Local Institution, Annāmalainagar
  - Local Institution, Bangalore
  - Local Institution, Chennai
  - Local Institution, Hyderabad
  - Local Institution, Indore
  - Local Institution, Kolkata
  - Local Institution, Kottayam
  - Local Institution, Lucknow
  - Local Institution, Mumbai Naka
  - Local Institution, Nashik
  - Local Institution, New Delhi
  - Local Institution, Pune
  - Local Institution, Thrissur
  - Local Institution, Vijayawada
- Israel (12):
  - Local Institution, Afula
  - Local Institution, Ashkelon
  - Local Institution, Giv‘atayim
  - Local Institution, Hadera
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Nazareth
  - Local Institution, Petah Tikva
  - Local Institution, Safed
  - Local Institution, Tel Aviv
- Italy (17):
  - Local Institution, Lido di Camaiore, Lucca
  - Local Institution, Ascoli Piceno
  - Local Institution, Campobasso
  - Local Institution, Chieti
  - Local Institution, Cremona
  - Local Institution, Fidenza (Pr)
  - Local Institution, Genova
  - Local Institution, Isernia
  - Local Institution, Livorno
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Palermo
  - Local Institution, Reggio Emilia
  - Local Institution, Roma
  - Local Institution, San Daniele de Friuli
  - Local Institution, Torino
  - Local Institution, Vittorio Veneto (Tv)
- Japan (41):
  - Local Institution, Itoshima, Fukuoka
  - Local Institution, Kurume, Fukuoka
  - Local Institution, Ohkawa-City, Fukuoka
  - Local Institution, Shirakawa, Fukushima
  - Local Institution, Takasaki, Gunma
  - Local Institution, Asahikawa-Shi, Hokkaido
  - Local Institution, Katou-Gun, Hokkaido
  - Local Institution, Katou-gun, Hokkaido
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Tomakomai-Shi, Hokkaido
  - Local Institution, Tomakomai-shi, Hokkaido
  - Local Institution, Yūbari, Hokkaido
  - Local Institution, Kobe, Hyōgo
  - Local Institution, Izumi, Kagoshima-ken
  - Local Institution, Isehara, Kanagawa
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Yokosuka, Kanagawa
  - Local Institution, Sendai, Miyagi
  - Local Institution, Nara, Nara
  - Local Institution, Izumi, Osaka
  - Local Institution, Osaka, Osaka
  - Local Institution, Suita, Osaka
  - Local Institution, Takatsuki, Osaka
  - Local Institution, Yao, Osaka
  - Local Institution, Saga, Saga-ken
  - Local Institution, Kasukabe-Shi, Saitama
  - Local Institution, Kasukabe-shi, Saitama
  - Local Institution, Itabashi-Ku, Tokyo
  - Local Institution, Itabashi-ku, Tokyo
  - Local Institution, Meguro-Ku, Tokyo
  - Local Institution, Meguro-ku, Tokyo
  - Local Institution, Shinagawa-Ku, Tokyo
  - Local Institution, Toyama, Toyama
  - Local Institution, Iwakuni, Yamaguchi
  - Local Institution, Fukui
  - Local Institution, Kagoshima
  - Local Institution, Kyoto
  - Local Institution, Nagasaki
  - Local Institution, Osaka
  - Local Institution, Ōita
  - Local Institution, Saga
- Malaysia (4):
  - Local Institution, Kubang Kerian, Kelantan
  - Local Institution, Kota Samarahan, Sarawak
  - Local Institution, Batu Caves, Selangor
  - Local Institution, Kuala Lumpur
- Mexico (10):
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Col. Toriello Guerra, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Morelia, Michoacán
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, Jalapa, Veracruz
  - Local Institution, Puebla City
  - Local Institution, Querétaro
- Netherlands (13):
  - Local Institution, 's-Hertogenbosch
  - Local Institution, Breda
  - Local Institution, Deventer
  - Local Institution, Eindhoven
  - Local Institution, Enschede
  - Local Institution, Hardenberg
  - Local Institution, Hilversum
  - Local Institution, Nijmegen
  - Local Institution, Oss
  - Local Institution, Rotterdam
  - Local Institution, Tiel
  - Local Institution, Utrecht
  - Local Institution, Velp
- Norway (11):
  - Local Institution, Ålesund
  - Local Institution, Bergen
  - Local Institution, Elverum
  - Local Institution, Flekkefjord
  - Local Institution, Nesttun
  - Local Institution, Oslo
  - Local Institution, Skien
  - Local Institution, Stavanger
  - Local Institution, Straume
  - Local Institution, Tromsø
  - Local Institution, Tønsberg
- Peru (7):
  - Local Institution, Chiclayo, Lambayeque
  - Local Institution, Jesus Maria, Lima region
  - Local Institution, Miraflores, Lima region
  - Local Institution, San Borja, Lima region
  - Local Institution, San Martín de Porres, Lima region
  - Local Institution, Bellavista, Provincia Constitucional del Callao
  - Local Institution, Lima
- Philippines (7):
  - Local Institution, Laoag, Ilocos Norte
  - Local Institution, Manila
  - Local Institution, Naga
  - Local Institution, Pasig
  - Local Institution, Quezon
  - Local Institution, Quezon City
  - Local Institution, San Juan City
- Poland (16):
  - Local Institution, Gdynia
  - Local Institution, Grodzisk Mazowiecki
  - Local Institution, Inowrocław
  - Local Institution, Kielce
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Piotrkow Trybunalski
  - Local Institution, Poznan
  - Local Institution, Płock
  - Local Institution, Płońsk
  - Local Institution, Ruda Śląska
  - Local Institution, Skierniewice
  - Local Institution, Słupsk
  - Local Institution, Torun
  - Local Institution, Warsaw
  - Local Institution, Węgrów
- Puerto Rico (3):
  - Local Institution, Cayey
  - Local Institution, Cidra
  - Local Institution, Ponce
- Romania (8):
  - Local Institution, Baia Mare
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
  - Local Institution, Iași
  - Local Institution, Oradea
  - Local Institution, Sibiu
  - Local Institution, Târgu Mureş
  - Local Institution, Timișoara
- Russia (25):
  - Local Institution, Chelyabinsk
  - Local Institution, Chita
  - Local Institution, Dzerzhinskiy
  - Local Institution, Kazan'
  - Local Institution, Kemerovo
  - Local Institution, Kirovsk
  - Local Institution, Krasnodar
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Novosibirsk
  - Local Institution, Odintsovo
  - Local Institution, Penza
  - Local Institution, Perm
  - Local Institution, Rostov-on-Don
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Saratov
  - Local Institution, Tomsk
  - Local Institution, Tver'
  - Local Institution, Tyumen
  - Local Institution, Voronezh
  - Local Institution, Yaroslavl
  - Local Institution, Zheleznodorozhniy
  - Local Institution, Zhukovsky
- Local Institution, Singapore, Singapore
- South Africa (9):
  - Local Institution, Westdene, Bloemfontein
  - Local Institution, Observatory, CAPE TOWN
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Richards Bay, KwaZulu-Natal
  - Local Institution, Bellville Cape Town, Western Cape
  - Local Institution, George, Western Cape
  - Local Institution, Parow, Western Cape
  - Local Institution, Somerset West, Western Cape
  - Local Institution, Worcester, Western Cape
- South Korea (12):
  - Local Institution, Anyang-si, Gyeonggi-do
  - Local Institution, Incheon, Korea
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Goyang
  - Local Institution, Gwangju
  - Local Institution, Gyeonggi-do
  - Local Institution, Pusan
  - Local Institution, Scongnam-Si
  - Local Institution, Seoul
  - Local Institution, Suwon
- Spain (15):
  - Local Institution, San Juan, Alicante
  - Local Institution, Torrevieja, Alicante
  - Local Institution, La Cañada, Almeria
  - Local Institution, Lugo, Galicia
  - Local Institution, Albacete
  - Local Institution, Barcelona
  - Local Institution, Elda
  - Local Institution, Figueres
  - Local Institution, Girona
  - Local Institution, Las Palmas
  - Local Institution, Madrid
  - Local Institution, Palma de Mallorca
  - Local Institution, San Sebastián de los Reyes
  - Local Institution, Tarragona
  - Local Institution, Viladecans
- Sweden (9):
  - Local Institution, Goteberg
  - Local Institution, Helsingborg
  - Local Institution, Linköping
  - Local Institution, Lund
  - Local Institution, Örebro
  - Local Institution, Skellefteå
  - Local Institution, Stockholm
  - Local Institution, Uppsala
  - Local Institution, Vaxjo
- Switzerland (2):
  - Local Institution, Baden
  - Local Institution, Bern
- Local Institution, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Local Institution, Ankara
  - Local Institution, Eskişehir
  - Local Institution, Izmir
- Ukraine (16):
  - Local Institution, Chernivtsy
  - Local Institution, Dnipropetrovsk
  - Local Institution, Donetsk
  - Local Institution, Ivano-Frankivsk
  - Local Institution, Kharkiv
  - Local Institution, Kiev
  - Local Institution, Kyiv
  - Local Institution, Luhansk
  - Local Institution, Lutsk
  - Local Institution, Lviv
  - Local Institution, Mykolayiv
  - Local Institution, Odesa
  - Local Institution, Uzhhorod
  - Local Institution, Vinnitsa
  - Local Institution, Zaporizhzhya
  - Local Institution, Zhytomyr
- United Kingdom (37):
  - Local Institution, Aberdeen, Aberdeenshire
  - Local Institution, Glasgow, Aberdeenshire
  - Local Institution, Belfast, Antrim
  - Local Institution, Craigavon, Armagh
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, Peterborough, Cambridgeshire
  - Local Institution, Chesterfield, Derbyshire
  - Local Institution, Bournemouth, Dorset
  - Local Institution, Glasgow, Dumbartonshire
  - Local Institution, Chichester, EAST Sussex
  - Local Institution, Colchester, Essex
  - Local Institution, Romford, Essex
  - Local Institution, Denmark Hill, Greater London
  - Local Institution, London, Greater London
  - Local Institution, Newport, Gwent
  - Local Institution, Barnet, Hertfordshire
  - Local Institution, Cardiff, MID Glamorgan
  - Local Institution, Llandough, MID Glamorgan
  - Local Institution, Harrow, Middlesex
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Worksop, Nottinghamshire
  - Local Institution, Paisley, Renfrewshire
  - Local Institution, Barnsley, South Yorkshire
  - Local Institution, Doncaster, South Yorkshire
  - Local Institution, Stirling, Stirlingshire
  - Local Institution, Glasgow, Strathclyde
  - Local Institution, Bury St Edmunds, Suffolk
  - Local Institution, Ipswich, Suffolk
  - Local Institution, Newcastle upon Tyne, TYNE and WEAR
  - Local Institution, Swansea, WEST Glamorgan
  - Local Institution, Livingston, WEST Lothian
  - Local Institution, Birmingham, WEST Midlands
  - Local Institution, Westbury, Wiltshire
  - Local Institution, York, Yorkshire
  - Local Institution, Antrim
  - Local Institution, Blackpool
  - Local Institution, Glasgow

REFERENCES:
- [Derived] Vinereanu D, Wojdyla DM, Alexander JH, Lopes RD, Al-Khatib SM, Gersh BJ, Bahit MC, Hohnloser SH, Flaker GC, Rosenquist M, Hijazi Z, Wallentin L, Granger CB. Heart rate and death and hospitalization for heart failure in patients with persistent or permanent atrial fibrillation: Insights from the ARISTOTLE trial. Am Heart J. 2023 Nov;265:132-136. doi: 10.1016/j.ahj.2023.07.006. Epub 2023 Jul 26. PMID 37506747
- [Derived] Hijazi Z, Lindback J, Oldgren J, Benz AP, Alexander JH, Connolly SJ, Eikelboom JW, Granger CB, Lopes RD, Siegbahn A, Wallentin L. Individual net clinical outcome with oral anticoagulation in atrial fibrillation using the ABC-AF risk scores. Am Heart J. 2023 Jul;261:55-63. doi: 10.1016/j.ahj.2023.03.012. Epub 2023 Mar 27. PMID 36990261
- [Derived] Jamieson MJ, Byon W, Dettloff RW, Crawford M, Gargalovic PS, Merali SJ, Onorato J, Quintero AJ, Russ C. Apixaban Use in Obese Patients: A Review of the Pharmacokinetic, Interventional, and Observational Study Data. Am J Cardiovasc Drugs. 2022 Nov;22(6):615-631. doi: 10.1007/s40256-022-00524-x. Epub 2022 May 16. PMID 35570249
- [Derived] Pol T, Hijazi Z, Lindback J, Oldgren J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Granger CB, Lopes RD, Yusuf S, Siegbahn A, Wallentin L. Using multimarker screening to identify biomarkers associated with cardiovascular death in patients with atrial fibrillation. Cardiovasc Res. 2022 Jul 20;118(9):2112-2123. doi: 10.1093/cvr/cvab262. PMID 34358298
- [Derived] Pol T, Hijazi Z, Lindback J, Alexander JH, Bahit MC, De Caterina R, Eikelboom JW, Ezekowitz MD, Gersh BJ, Granger CB, Hylek EM, Lopes R, Siegbahn A, Wallentin L. Evaluation of the prognostic value of GDF-15, ABC-AF-bleeding score and ABC-AF-death score in patients with atrial fibrillation across different geographical areas. Open Heart. 2021 Mar;8(1):e001471. doi: 10.1136/openhrt-2020-001471. PMID 33741689
- [Derived] Hijazi Z, Wallentin L, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Granger CB, Lopes RD, Pol T, Yusuf S, Oldgren J, Siegbahn A. Screening of Multiple Biomarkers Associated With Ischemic Stroke in Atrial Fibrillation. J Am Heart Assoc. 2020 Dec 15;9(24):e018984. doi: 10.1161/JAHA.120.018984. Epub 2020 Dec 9. PMID 33292046
- [Derived] Wallentin L, Lindback J, Eriksson N, Hijazi Z, Eikelboom JW, Ezekowitz MD, Granger CB, Lopes RD, Yusuf S, Oldgren J, Siegbahn A. Angiotensin-converting enzyme 2 (ACE2) levels in relation to risk factors for COVID-19 in two large cohorts of patients with atrial fibrillation. Eur Heart J. 2020 Nov 1;41(41):4037-4046. doi: 10.1093/eurheartj/ehaa697. PMID 32984892
- [Derived] Hijazi Z, Granger CB, Hohnloser SH, Westerbergh J, Lindback J, Alexander JH, Keltai M, Parkhomenko A, Lopez-Sendon JL, Lopes RD, Siegbahn A, Wallentin L. Association of Different Estimates of Renal Function With Cardiovascular Mortality and Bleeding in Atrial Fibrillation. J Am Heart Assoc. 2020 Sep 15;9(18):e017155. doi: 10.1161/JAHA.120.017155. Epub 2020 Aug 31. PMID 32865097
- [Derived] Zeitouni M, Giczewska A, Alexander JH. Reply: Specifics of Dose Modification in ARISTOTLE. J Am Coll Cardiol. 2020 Jul 7;76(1):128-129. doi: 10.1016/j.jacc.2020.05.013. No abstract available. PMID 32616154
- [Derived] Rosjo H, Hijazi Z, Omland T, Westerbergh J, Lyngbakken MN, Alexander JH, Gersh BJ, Granger CB, Hylek EM, Lopes RD, Siegbahn A, Wallentin L. Cardiac troponin is associated with cardiac outcomes in men and women with atrial fibrillation, insights from the ARISTOTLE trial. J Intern Med. 2020 Aug;288(2):248-259. doi: 10.1111/joim.13072. Epub 2020 May 18. PMID 32350915
- [Derived] Zeitouni M, Giczewska A, Lopes RD, Wojdyla DM, Christersson C, Siegbahn A, De Caterina R, Steg PG, Granger CB, Wallentin L, Alexander JH; ARISTOTLE Investigators. Clinical and Pharmacological Effects of Apixaban Dose Adjustment in the ARISTOTLE Trial. J Am Coll Cardiol. 2020 Mar 17;75(10):1145-1155. doi: 10.1016/j.jacc.2019.12.060. PMID 32164888
- [Derived] Stanifer JW, Pokorney SD, Chertow GM, Hohnloser SH, Wojdyla DM, Garonzik S, Byon W, Hijazi Z, Lopes RD, Alexander JH, Wallentin L, Granger CB. Apixaban Versus Warfarin in Patients With Atrial Fibrillation and Advanced Chronic Kidney Disease. Circulation. 2020 Apr 28;141(17):1384-1392. doi: 10.1161/CIRCULATIONAHA.119.044059. Epub 2020 Mar 12. PMID 32160801
- [Derived] Garcia DA, Fisher DA, Mulder H, Wruck L, De Caterina R, Halvorsen S, Granger CB, Held C, Wallentin L, Alexander JH, Lopes RD. Gastrointestinal bleeding in patients with atrial fibrillation treated with Apixaban or warfarin: Insights from the Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) trial. Am Heart J. 2020 Mar;221:1-8. doi: 10.1016/j.ahj.2019.10.013. Epub 2019 Oct 31. PMID 31896036
- [Derived] Dalgaard F, Mulder H, Wojdyla DM, Lopes RD, Held C, Alexander JH, De Caterina R, Washam JB, Hylek EM, Garcia DA, Gersh BJ, Wallentin L, Granger CB, Al-Khatib SM. Patients With Atrial Fibrillation Taking Nonsteroidal Anti-Inflammatory Drugs and Oral Anticoagulants in the ARISTOTLE Trial. Circulation. 2020 Jan 7;141(1):10-20. doi: 10.1161/CIRCULATIONAHA.119.041296. Epub 2019 Nov 21. PMID 31747786
- [Derived] Goldstein SA, Green J, Huber K, Wojdyla DM, Lopes RD, Alexander JH, Vinereanu D, Wallentin L, Granger CB, Al-Khatib SM. Characteristics and Outcomes of Atrial Fibrillation in Patients With Thyroid Disease (from the ARISTOTLE Trial). Am J Cardiol. 2019 Nov 1;124(9):1406-1412. doi: 10.1016/j.amjcard.2019.07.046. Epub 2019 Aug 7. PMID 31474328
- [Derived] Guimaraes PO, Pokorney SD, Lopes RD, Wojdyla DM, Gersh BJ, Giczewska A, Carnicelli A, Lewis BS, Hanna M, Wallentin L, Vinereanu D, Alexander JH, Granger CB. Efficacy and safety of apixaban vs warfarin in patients with atrial fibrillation and prior bioprosthetic valve replacement or valve repair: Insights from the ARISTOTLE trial. Clin Cardiol. 2019 May;42(5):568-571. doi: 10.1002/clc.23178. Epub 2019 Apr 9. PMID 30907005
- [Derived] Washam JB, Hohnloser SH, Lopes RD, Wojdyla DM, Vinereanu D, Alexander JH, Gersh BJ, Hanna M, Horowitz J, Hylek EM, Xavier D, Verheugt FWA, Wallentin L, Granger CB; ARISTOTLE Committees and Investigators. Interacting medication use and the treatment effects of apixaban versus warfarin: results from the ARISTOTLE Trial. J Thromb Thrombolysis. 2019 Apr;47(3):345-352. doi: 10.1007/s11239-019-01823-y. PMID 30790160
- [Derived] Hohnloser SH, Fudim M, Alexander JH, Wojdyla DM, Ezekowitz JA, Hanna M, Atar D, Hijazi Z, Bahit MC, Al-Khatib SM, Lopez-Sendon JL, Wallentin L, Granger CB, Lopes RD. Efficacy and Safety of Apixaban Versus Warfarin in Patients With Atrial Fibrillation and Extremes in Body Weight. Circulation. 2019 May 14;139(20):2292-2300. doi: 10.1161/CIRCULATIONAHA.118.037955. PMID 30773022
- [Derived] Alexander KP, Brouwer MA, Mulder H, Vinereanu D, Lopes RD, Proietti M, Al-Khatib SM, Hijazi Z, Halvorsen S, Hylek EM, Verheugt FWA, Alexander JH, Wallentin L, Granger CB; ARISTOTLE Investigators. Outcomes of apixaban versus warfarin in patients with atrial fibrillation and multi-morbidity: Insights from the ARISTOTLE trial. Am Heart J. 2019 Feb;208:123-131. doi: 10.1016/j.ahj.2018.09.017. Epub 2018 Nov 22. PMID 30579505
- [Derived] Sandhu RK, Ezekowitz JA, Hijazi Z, Westerbergh J, Aulin J, Alexander JH, Granger CB, Halvorsen S, Hanna MS, Lopes RD, Siegbahn A, Wallentin L. Obesity paradox on outcome in atrial fibrillation maintained even considering the prognostic influence of biomarkers: insights from the ARISTOTLE trial. Open Heart. 2018 Nov 1;5(2):e000908. doi: 10.1136/openhrt-2018-000908. eCollection 2018. PMID 30487982
- [Derived] Christersson C, Wallentin L, Andersson U, Alexander JH, Alings M, De Caterina R, Gersh BJ, Granger CB, Halvorsen S, Hanna M, Huber K, Hylek EM, Lopes RD, Oh BH, Siegbahn A. Effect of apixaban compared with warfarin on coagulation markers in atrial fibrillation. Heart. 2019 Feb;105(3):235-242. doi: 10.1136/heartjnl-2018-313351. Epub 2018 Sep 12. PMID 30209126
- [Derived] Horowitz JD, De Caterina R, Heresztyn T, Alexander JH, Andersson U, Lopes RD, Steg PG, Hylek EM, Mohan P, Hanna M, Jansky P, Granger CB, Wallentin L; ARISTOTLE Investigators. Asymmetric and Symmetric Dimethylarginine Predict Outcomes in Patients With Atrial Fibrillation: An ARISTOTLE Substudy. J Am Coll Cardiol. 2018 Aug 14;72(7):721-733. doi: 10.1016/j.jacc.2018.05.058. PMID 30092948
- [Derived] Sharma A, Hijazi Z, Andersson U, Al-Khatib SM, Lopes RD, Alexander JH, Held C, Hylek EM, Leonardi S, Hanna M, Ezekowitz JA, Siegbahn A, Granger CB, Wallentin L. Use of Biomarkers to Predict Specific Causes of Death in Patients With Atrial Fibrillation. Circulation. 2018 Oct 16;138(16):1666-1676. doi: 10.1161/CIRCULATIONAHA.118.034125. PMID 29871978
- [Derived] Kopin D, Jones WS, Sherwood MW, Wojdyla DM, Wallentin L, Lewis BS, Verheugt FWA, Vinereanu D, Bahit MC, Halvorsen S, Huber K, Parkhomenko A, Granger CB, Lopes RD, Alexander JH. Percutaneous coronary intervention and antiplatelet therapy in patients with atrial fibrillation receiving apixaban or warfarin: Insights from the ARISTOTLE trial. Am Heart J. 2018 Mar;197:133-141. doi: 10.1016/j.ahj.2017.11.005. Epub 2017 Nov 10. PMID 29447773
- [Derived] Pol T, Held C, Westerbergh J, Lindback J, Alexander JH, Alings M, Erol C, Goto S, Halvorsen S, Huber K, Hanna M, Lopes RD, Ruzyllo W, Granger CB, Hijazi Z. Dyslipidemia and Risk of Cardiovascular Events in Patients With Atrial Fibrillation Treated With Oral Anticoagulation Therapy: Insights From the ARISTOTLE (Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation) Trial. J Am Heart Assoc. 2018 Feb 1;7(3):e007444. doi: 10.1161/JAHA.117.007444. PMID 29419390
- [Derived] Goto S, Merrill P, Wallentin L, Wojdyla DM, Hanna M, Avezum A, Easton JD, Harjola VP, Huber K, Lewis BS, Parkhomenko A, Zhu J, Granger CB, Lopes RD, Alexander JH. Antithrombotic therapy use and clinical outcomes following thrombo-embolic events in patients with atrial fibrillation: insights from ARISTOTLE. Eur Heart J Cardiovasc Pharmacother. 2018 Apr 1;4(2):75-81. doi: 10.1093/ehjcvp/pvy002. PMID 29385429
- [Derived] Vinereanu D, Wang A, Mulder H, Lopes RD, Jansky P, Lewis BS, Gersh BJ, Avezum A, Hanna M, Held C, Wallentin L, Granger CB, Alexander JH. Outcomes in anticoagulated patients with atrial fibrillation and with mitral or aortic valve disease. Heart. 2018 Aug;104(15):1292-1299. doi: 10.1136/heartjnl-2017-312272. Epub 2018 Jan 19. PMID 29352007
- [Derived] Rao MP, Vinereanu D, Wojdyla DM, Alexander JH, Atar D, Hylek EM, Hanna M, Wallentin L, Lopes RD, Gersh BJ, Granger CB; Apixaban for Reduction in Stroke Other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) Investigators. Clinical Outcomes and History of Fall in Patients with Atrial Fibrillation Treated with Oral Anticoagulation: Insights From the ARISTOTLE Trial. Am J Med. 2018 Mar;131(3):269-275.e2. doi: 10.1016/j.amjmed.2017.10.036. Epub 2017 Nov 6. PMID 29122636
- [Derived] Vinereanu D, Lopes RD, Mulder H, Gersh BJ, Hanna M, de Barros E Silva PGM, Atar D, Wallentin L, Granger CB, Alexander JH; ARISTOTLE Investigators. Echocardiographic Risk Factors for Stroke and Outcomes in Patients With Atrial Fibrillation Anticoagulated With Apixaban or Warfarin. Stroke. 2017 Dec;48(12):3266-3273. doi: 10.1161/STROKEAHA.117.017574. Epub 2017 Oct 31. PMID 29089455
- [Derived] Hijazi Z, Oldgren J, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Held C, Hylek EM, Lopes RD, Yusuf S, Granger CB, Siegbahn A, Wallentin L; ARISTOTLE and RE-LY Investigators. A biomarker-based risk score to predict death in patients with atrial fibrillation: the ABC (age, biomarkers, clinical history) death risk score. Eur Heart J. 2018 Feb 7;39(6):477-485. doi: 10.1093/eurheartj/ehx584. PMID 29069359
- [Derived] Hijazi Z, Lindahl B, Oldgren J, Andersson U, Lindback J, Granger CB, Alexander JH, Gersh BJ, Hanna M, Harjola VP, Hylek EM, Lopes RD, Siegbahn A, Wallentin L. Repeated Measurements of Cardiac Biomarkers in Atrial Fibrillation and Validation of the ABC Stroke Score Over Time. J Am Heart Assoc. 2017 Jun 23;6(6):e004851. doi: 10.1161/JAHA.116.004851. PMID 28645934
- [Derived] Lopes RD, Guimaraes PO, Kolls BJ, Wojdyla DM, Bushnell CD, Hanna M, Easton JD, Thomas L, Wallentin L, Al-Khatib SM, Held C, Gabriel Melo de Barros E Silva P, Alexander JH, Granger CB, Diener HC. Intracranial hemorrhage in patients with atrial fibrillation receiving anticoagulation therapy. Blood. 2017 Jun 1;129(22):2980-2987. doi: 10.1182/blood-2016-08-731638. Epub 2017 Mar 29. PMID 28356246
- [Derived] Cowper PA, Sheng S, Lopes RD, Anstrom KJ, Stafford JA, Davidson-Ray L, Al-Khatib SM, Ansell J, Dorian P, Husted S, McMurray JJV, Steg PG, Alexander JH, Wallentin L, Granger CB, Mark DB. Economic Analysis of Apixaban Therapy for Patients With Atrial Fibrillation From a US Perspective: Results From the ARISTOTLE Randomized Clinical Trial. JAMA Cardiol. 2017 May 1;2(5):525-534. doi: 10.1001/jamacardio.2017.0065. PMID 28355434
- [Derived] Hu PT, Lopes RD, Stevens SR, Wallentin L, Thomas L, Alexander JH, Hanna M, Lewis BS, Verheugt FW, Granger CB, Jones WS. Efficacy and Safety of Apixaban Compared With Warfarin in Patients With Atrial Fibrillation and Peripheral Artery Disease: Insights From the ARISTOTLE Trial. J Am Heart Assoc. 2017 Jan 17;6(1):e004699. doi: 10.1161/JAHA.116.004699. PMID 28096100
- [Derived] Bahit MC, Lopes RD, Wojdyla DM, Held C, Hanna M, Vinereanu D, Hylek EM, Verheugt F, Goto S, Alexander JH, Wallentin L, Granger CB. Non-major bleeding with apixaban versus warfarin in patients with atrial fibrillation. Heart. 2017 Apr;103(8):623-628. doi: 10.1136/heartjnl-2016-309901. Epub 2016 Oct 24. PMID 27798052
- [Derived] Oldgren J, Hijazi Z, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Granger CB, Hylek EM, Lopes RD, Siegbahn A, Yusuf S, Wallentin L; RE-LY and ARISTOTLE Investigators. Performance and Validation of a Novel Biomarker-Based Stroke Risk Score for Atrial Fibrillation. Circulation. 2016 Nov 29;134(22):1697-1707. doi: 10.1161/CIRCULATIONAHA.116.022802. Epub 2016 Aug 28. PMID 27569438
- [Derived] Alexander JH, Andersson U, Lopes RD, Hijazi Z, Hohnloser SH, Ezekowitz JA, Halvorsen S, Hanna M, Commerford P, Ruzyllo W, Huber K, Al-Khatib SM, Granger CB, Wallentin L; Apixaban for Reduction of Stroke and Other Thromboembolic Complications in Atrial Fibrillation (ARISTOTLE) Investigators. Apixaban 5 mg Twice Daily and Clinical Outcomes in Patients With Atrial Fibrillation and Advanced Age, Low Body Weight, or High Creatinine: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2016 Sep 1;1(6):673-81. doi: 10.1001/jamacardio.2016.1829. PMID 27463942
- [Derived] Hijazi Z, Hohnloser SH, Andersson U, Alexander JH, Hanna M, Keltai M, Parkhomenko A, Lopez-Sendon JL, Lopes RD, Siegbahn A, Granger CB, Wallentin L. Efficacy and Safety of Apixaban Compared With Warfarin in Patients With Atrial Fibrillation in Relation to Renal Function Over Time: Insights From the ARISTOTLE Randomized Clinical Trial. JAMA Cardiol. 2016 Jul 1;1(4):451-60. doi: 10.1001/jamacardio.2016.1170. PMID 27438322
- [Derived] Jaspers Focks J, Brouwer MA, Wojdyla DM, Thomas L, Lopes RD, Washam JB, Lanas F, Xavier D, Husted S, Wallentin L, Alexander JH, Granger CB, Verheugt FW. Polypharmacy and effects of apixaban versus warfarin in patients with atrial fibrillation: post hoc analysis of the ARISTOTLE trial. BMJ. 2016 Jun 15;353:i2868. doi: 10.1136/bmj.i2868. PMID 27306620
- [Derived] Hijazi Z, Oldgren J, Lindback J, Alexander JH, Connolly SJ, Eikelboom JW, Ezekowitz MD, Held C, Hylek EM, Lopes RD, Siegbahn A, Yusuf S, Granger CB, Wallentin L; ARISTOTLE and RE-LY Investigators. The novel biomarker-based ABC (age, biomarkers, clinical history)-bleeding risk score for patients with atrial fibrillation: a derivation and validation study. Lancet. 2016 Jun 4;387(10035):2302-2311. doi: 10.1016/S0140-6736(16)00741-8. Epub 2016 Apr 4. PMID 27056738
- [Derived] Hijazi Z, Lindback J, Alexander JH, Hanna M, Held C, Hylek EM, Lopes RD, Oldgren J, Siegbahn A, Stewart RA, White HD, Granger CB, Wallentin L; ARISTOTLE and STABILITY Investigators. The ABC (age, biomarkers, clinical history) stroke risk score: a biomarker-based risk score for predicting stroke in atrial fibrillation. Eur Heart J. 2016 May 21;37(20):1582-90. doi: 10.1093/eurheartj/ehw054. Epub 2016 Feb 25. PMID 26920728
- [Derived] Hijazi Z, Aulin J, Andersson U, Alexander JH, Gersh B, Granger CB, Hanna M, Horowitz J, Hylek EM, Lopes RD, Siegbahn A, Wallentin L; ARISTOTLE Investigators. Biomarkers of inflammation and risk of cardiovascular events in anticoagulated patients with atrial fibrillation. Heart. 2016 Apr;102(7):508-17. doi: 10.1136/heartjnl-2015-308887. Epub 2016 Feb 2. PMID 26839066
- [Derived] Rao MP, Halvorsen S, Wojdyla D, Thomas L, Alexander JH, Hylek EM, Hanna M, Bahit MC, Lopes RD, De Caterina R, Erol C, Goto S, Lanas F, Lewis BS, Husted S, Gersh BJ, Wallentin L, Granger CB; Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) Steering Committee and Investigators. Blood Pressure Control and Risk of Stroke or Systemic Embolism in Patients With Atrial Fibrillation: Results From the Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) Trial. J Am Heart Assoc. 2015 Dec 1;4(12):e002015. doi: 10.1161/JAHA.115.002015. PMID 26627878
- [Derived] Vinereanu D, Stevens SR, Alexander JH, Al-Khatib SM, Avezum A, Bahit MC, Granger CB, Lopes RD, Halvorsen S, Hanna M, Husted S, Hylek EM, Margulescu AD, Wallentin L, Atar D. Clinical outcomes in patients with atrial fibrillation according to sex during anticoagulation with apixaban or warfarin: a secondary analysis of a randomized controlled trial. Eur Heart J. 2015 Dec 7;36(46):3268-75. doi: 10.1093/eurheartj/ehv447. Epub 2015 Sep 14. PMID 26371113
- [Derived] Avezum A, Lopes RD, Schulte PJ, Lanas F, Gersh BJ, Hanna M, Pais P, Erol C, Diaz R, Bahit MC, Bartunek J, De Caterina R, Goto S, Ruzyllo W, Zhu J, Granger CB, Alexander JH. Apixaban in Comparison With Warfarin in Patients With Atrial Fibrillation and Valvular Heart Disease: Findings From the Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) Trial. Circulation. 2015 Aug 25;132(8):624-32. doi: 10.1161/CIRCULATIONAHA.114.014807. Epub 2015 Jun 23. PMID 26106009
- [Derived] Held C, Hylek EM, Alexander JH, Hanna M, Lopes RD, Wojdyla DM, Thomas L, Al-Khalidi H, Alings M, Xavier D, Ansell J, Goto S, Ruzyllo W, Rosenqvist M, Verheugt FW, Zhu J, Granger CB, Wallentin L. Clinical outcomes and management associated with major bleeding in patients with atrial fibrillation treated with apixaban or warfarin: insights from the ARISTOTLE trial. Eur Heart J. 2015 May 21;36(20):1264-72. doi: 10.1093/eurheartj/ehu463. Epub 2014 Dec 12. PMID 25499871
- [Derived] Hijazi Z, Siegbahn A, Andersson U, Lindahl B, Granger CB, Alexander JH, Atar D, Gersh BJ, Hanna M, Harjola VP, Horowitz J, Husted S, Hylek EM, Lopes RD, McMurray JJ, Wallentin L. Comparison of cardiac troponins I and T measured with high-sensitivity methods for evaluation of prognosis in atrial fibrillation: an ARISTOTLE substudy. Clin Chem. 2015 Feb;61(2):368-78. doi: 10.1373/clinchem.2014.226936. Epub 2014 Dec 1. PMID 25451868
- [Derived] Garcia D, Alexander JH, Wallentin L, Wojdyla DM, Thomas L, Hanna M, Al-Khatib SM, Dorian P, Ansell J, Commerford P, Flaker G, Lanas F, Vinereanu D, Xavier D, Hylek EM, Held C, Verheugt FW, Granger CB, Lopes RD. Management and clinical outcomes in patients treated with apixaban vs warfarin undergoing procedures. Blood. 2014 Dec 11;124(25):3692-8. doi: 10.1182/blood-2014-08-595496. Epub 2014 Oct 15. PMID 25320240
- [Derived] Wallentin L, Hijazi Z, Andersson U, Alexander JH, De Caterina R, Hanna M, Horowitz JD, Hylek EM, Lopes RD, Asberg S, Granger CB, Siegbahn A; ARISTOTLE Investigators. Growth differentiation factor 15, a marker of oxidative stress and inflammation, for risk assessment in patients with atrial fibrillation: insights from the Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) trial. Circulation. 2014 Nov 18;130(21):1847-58. doi: 10.1161/CIRCULATIONAHA.114.011204. Epub 2014 Oct 7. PMID 25294786
- [Derived] Hijazi Z, Siegbahn A, Andersson U, Granger CB, Alexander JH, Atar D, Gersh BJ, Mohan P, Harjola VP, Horowitz J, Husted S, Hylek EM, Lopes RD, McMurray JJ, Wallentin L; ARISTOTLE Investigators. High-sensitivity troponin I for risk assessment in patients with atrial fibrillation: insights from the Apixaban for Reduction in Stroke and other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) trial. Circulation. 2014 Feb 11;129(6):625-34. doi: 10.1161/CIRCULATIONAHA.113.006286. Epub 2013 Nov 13. PMID 24226808
- [Derived] Flaker G, Lopes RD, Al-Khatib SM, Hermosillo AG, Hohnloser SH, Tinga B, Zhu J, Mohan P, Garcia D, Bartunek J, Vinereanu D, Husted S, Harjola VP, Rosenqvist M, Alexander JH, Granger CB; ARISTOTLE Committees and Investigators. Efficacy and safety of apixaban in patients after cardioversion for atrial fibrillation: insights from the ARISTOTLE Trial (Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation). J Am Coll Cardiol. 2014 Mar 25;63(11):1082-7. doi: 10.1016/j.jacc.2013.09.062. Epub 2013 Nov 6. PMID 24211508
- [Derived] Hijazi Z, Wallentin L, Siegbahn A, Andersson U, Alexander JH, Atar D, Gersh BJ, Hanna M, Harjola VP, Horowitz JD, Husted S, Hylek EM, Lopes RD, McMurray JJ, Granger CB; ARISTOTLE Investigators. High-sensitivity troponin T and risk stratification in patients with atrial fibrillation during treatment with apixaban or warfarin. J Am Coll Cardiol. 2014 Jan 7-14;63(1):52-61. doi: 10.1016/j.jacc.2013.07.093. Epub 2013 Sep 19. PMID 24055845
- [Derived] Alexander JH, Levy E, Lawrence J, Hanna M, Waclawski AP, Wang J, Califf RM, Wallentin L, Granger CB. Documentation of study medication dispensing in a prospective large randomized clinical trial: experiences from the ARISTOTLE Trial. Am Heart J. 2013 Sep;166(3):559-65. doi: 10.1016/j.ahj.2013.05.025. Epub 2013 Aug 15. PMID 24016507
- [Derived] Garcia DA, Wallentin L, Lopes RD, Thomas L, Alexander JH, Hylek EM, Ansell J, Hanna M, Lanas F, Flaker G, Commerford P, Xavier D, Vinereanu D, Yang H, Granger CB. Apixaban versus warfarin in patients with atrial fibrillation according to prior warfarin use: results from the Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation trial. Am Heart J. 2013 Sep;166(3):549-58. doi: 10.1016/j.ahj.2013.05.016. Epub 2013 Jul 25. PMID 24016506
- [Derived] Wallentin L, Lopes RD, Hanna M, Thomas L, Hellkamp A, Nepal S, Hylek EM, Al-Khatib SM, Alexander JH, Alings M, Amerena J, Ansell J, Aylward P, Bartunek J, Commerford P, De Caterina R, Erol C, Harjola VP, Held C, Horowitz JD, Huber K, Husted S, Keltai M, Lanas F, Lisheng L, McMurray JJ, Oh BH, Rosenqvist M, Ruzyllo W, Steg PG, Vinereanu D, Xavier D, Granger CB; Apixaban for Reduction in Stroke and Other Thromboembolic Events in Atrial Fibrillation (ARISTOTLE) Investigators. Efficacy and safety of apixaban compared with warfarin at different levels of predicted international normalized ratio control for stroke prevention in atrial fibrillation. Circulation. 2013 Jun 4;127(22):2166-76. doi: 10.1161/CIRCULATIONAHA.112.142158. Epub 2013 May 2. PMID 23640971
- [Derived] McMurray JJ, Ezekowitz JA, Lewis BS, Gersh BJ, van Diepen S, Amerena J, Bartunek J, Commerford P, Oh BH, Harjola VP, Al-Khatib SM, Hanna M, Alexander JH, Lopes RD, Wojdyla DM, Wallentin L, Granger CB; ARISTOTLE Committees and Investigators. Left ventricular systolic dysfunction, heart failure, and the risk of stroke and systemic embolism in patients with atrial fibrillation: insights from the ARISTOTLE trial. Circ Heart Fail. 2013 May;6(3):451-60. doi: 10.1161/CIRCHEARTFAILURE.112.000143. Epub 2013 Apr 10. PMID 23575255
- [Derived] Hijazi Z, Wallentin L, Siegbahn A, Andersson U, Christersson C, Ezekowitz J, Gersh BJ, Hanna M, Hohnloser S, Horowitz J, Huber K, Hylek EM, Lopes RD, McMurray JJ, Granger CB. N-terminal pro-B-type natriuretic peptide for risk assessment in patients with atrial fibrillation: insights from the ARISTOTLE Trial (Apixaban for the Prevention of Stroke in Subjects With Atrial Fibrillation). J Am Coll Cardiol. 2013 Jun 4;61(22):2274-84. doi: 10.1016/j.jacc.2012.11.082. Epub 2013 Apr 3. PMID 23563134
- [Derived] Lopes RD, Al-Khatib SM, Wallentin L, Yang H, Ansell J, Bahit MC, De Caterina R, Dorian P, Easton JD, Erol C, Ezekowitz JA, Gersh BJ, Granger CB, Hohnloser SH, Horowitz J, Hylek EM, McMurray JJ, Mohan P, Vinereanu D, Alexander JH. Efficacy and safety of apixaban compared with warfarin according to patient risk of stroke and of bleeding in atrial fibrillation: a secondary analysis of a randomised controlled trial. Lancet. 2012 Nov 17;380(9855):1749-58. doi: 10.1016/S0140-6736(12)60986-6. Epub 2012 Oct 2. PMID 23036896
- [Derived] Easton JD, Lopes RD, Bahit MC, Wojdyla DM, Granger CB, Wallentin L, Alings M, Goto S, Lewis BS, Rosenqvist M, Hanna M, Mohan P, Alexander JH, Diener HC; ARISTOTLE Committees and Investigators. Apixaban compared with warfarin in patients with atrial fibrillation and previous stroke or transient ischaemic attack: a subgroup analysis of the ARISTOTLE trial. Lancet Neurol. 2012 Jun;11(6):503-11. doi: 10.1016/S1474-4422(12)70092-3. Epub 2012 May 8. PMID 22572202
- [Derived] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20998 participants were enrolled, and 18201 were randomized.
Groups:
- Apixaban: Participants received apixaban and warfarin-placebo following randomization during a titration phase using a dosing algorithm for warfarin- placebo; apixaban was dosed at 5 mg twice daily (BID) [or 2.5 mg BID in select subjects]. Subsequent warfarin placebo doses were recommended based upon an algorithm using an encrypted, shammed International Normalized Ratio (INR) procedure to preserve the double blind; however, the final dosing decision rested with the investigator.
- Warfarin: Participants received apixaban-placebo and warfarin following randomization during a titration phase using a dosing algorithm for warfarin; apixaban-placebo was dosed at 5 mg twice daily (BID) [or 2.5 mg BID in select subjects]. Subsequent warfarin doses were recommended based upon an algorithm and encrypted INR testing to preserve the double blind; however, the final dosing decision rested with the investigator.
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 9120 (Randomized participants) | 9081 (Randomized participants)
Completed | 6810 | 6588
Not Completed | 2310 | 2493
Not completed — Death | 331 | 349
Not completed — Adverse Event | 679 | 738
Not completed — Withdrawal by Subject | 921 | 989
Not completed — Lost to Follow-up | 51 | 39
Not completed — Poor/Noncompliance | 57 | 77
Not completed — Pregnancy | 1 | 0
Not completed — Subject No Longer Meets Study Criteria | 87 | 100
Not completed — Administrative Reason by Sponsor | 11 | 8
Not completed — Physician Refused to Continue Treatment | 81 | 89
Not completed — Other Reason | 80 | 92
Not completed — Not Reported | 11 | 12

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 9120 | 9081 | 18201
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.61) | 69.0 (9.74) | 69.1 (9.68)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 2731 | 2740 | 5471
  Between 65 and 75 years | 3539 | 3513 | 7052
  >=75 years | 2850 | 2828 | 5678
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3234 | 3182 | 6416
  Male | 5886 | 5899 | 11785
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White (European) | 5440 | 5366 | 10806
  White (Middle Eastern or North African) | 59 | 66 | 125
  White (Other White) | 2037 | 2060 | 4097
  White (Not Reported) | 0 | 1 | 1
  Black / African American | 125 | 102 | 227
  Asian (Asian Indian) | 307 | 312 | 619
  Asian (Chinese) | 536 | 536 | 1072
  Asian (Japanese) | 164 | 180 | 344
  Asian (Other Asian) | 303 | 304 | 607
  American Indian / Alaska Native | 26 | 24 | 50
  Native Hawaiian / Other Pacific Islander | 2 | 2 | 4
  Other | 121 | 127 | 248
  Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic / Latino | 1808 | 1803 | 3611
  Not Hispanic / Latino | 7312 | 7276 | 14588
  Not Reported | 0 | 2 | 2
Female Age Category [Count of Participants; unit: Participants]
  <=50 years | 81 | 88 | 169
  >50 years | 3153 | 3094 | 6247
  not applicable (male) | 5886 | 5899 | 11785
Apixaban/Matching Placebo Dose at Randomization [Count of Participants; unit: Participants]
  2.5 mg twice daily (BID) | 428 | 403 | 831
  5.0 mg BID | 8692 | 8678 | 17370
Risk Factor at Enrollment: Age >= 75 Years [Count of Participants; unit: Participants]
  >=75 years | 2850 | 2828 | 5678
  <75 years | 6270 | 6253 | 12523
Risk Factor at Enrollment: Prior Stroke [Count of Participants; unit: Participants]
  With prior stroke | 1045 | 1082 | 2127
  Prior stroke not a risk factor | 8075 | 7999 | 16074
Risk Factor at Enrollment: Prior Transient Ischemic Attack (TIA) [Count of Participants; unit: Participants]
  With prior TIA | 603 | 654 | 1257
  Prior TIA not a risk factor | 8517 | 8427 | 16944
Risk Factor At Enrollment: Symptomatic Chronic Heart Failure (CHF) [Count of Participants; unit: Participants]
  With symptomatic CHF | 2784 | 2757 | 5541
  Symptomatic CHF not a risk factor | 6336 | 6324 | 12660
Risk Factor at Enrollment: Left Ventricle Ejection Fraction (LVEF) <=40% [Count of Participants; unit: Participants]
  With LVEF <=40% | 1324 | 1301 | 2625
  LVEF <=40% not a risk factor | 7796 | 7780 | 15576
Number of Risk Factors [Count of Participants; unit: Participants]
  <= 1 | 3025 | 3000 | 6025
  >= 2 | 6095 | 6081 | 12176
CHADS-2 Score at Enrollment [Count of Participants; unit: Participants] — The CHADS2 score is a clinical prediction rule for estimating the risk of stroke in patients with nonrheumatic atrial fibrillation (AF). A high CHADS2 score corresponds to a greater risk of stroke, while a low CHADS2 score corresponds to a lower risk of stroke (range 0 to 6). The CHADS2 score is determined by adding together the points that correspond to the 5 conditions that are present: 1 point each for congestive heart failure, hypertension, age ≥75 years, or diabetes mellitus; 2 points for prior stroke or transient ischemic attack (TIA).
  Participants
    Score of <= 1 | 3100 | 3083 | 6183
    Score of 2 | 3262 | 3254 | 6516
    Score of >= 3 | 2758 | 2744 | 5502
Mean CHADS-2 Score at Enrollment [Mean (Standard Deviation); unit: units on a scale] — The CHADS2 score is a clinical prediction rule for estimating the risk of stroke in patients with nonrheumatic atrial fibrillation (AF). A high CHADS2 score corresponds to a greater risk of stroke, while a low CHADS2 score corresponds to a lower risk of stroke (range 0 to 6). The CHADS2 score is determined by adding together the points that correspond to the 5 conditions that are present: 1 point each for Congestive Heart Failure, Hypertension, Age ≥75 years, or Diabetes Mellitus; 2 points for prior stroke or transient ischemic attack (TIA).
  units on a scale | 2.1 (1.10) | 2.1 (1.11) | 2.1 (2.10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Event of Ischemic/Unspecified Stroke, Hemorrhagic Stroke, or Systemic Embolism (SE) During the Intended Treatment Period
Description: All suspected efficacy events were adjudicated by the Central Events Committee (CEC). Diagnosis of stroke=the nontraumatic focal neurological deficit lasting at least 24 hours, and includes ischemic stroke, hemorrhagic stroke, ischemic stroke with hemorrhagic conversion, stroke of uncertain type, and retinal ischemic event (embolism, infarction). Diagnosis of SE=clinical history consistent with an acute loss of blood flow to a peripheral artery (or arteries), supported by evidence of embolism from surgical specimens, autopsy, angiography, vascular imaging, or other objective testing.
Time Frame: Time to first event in "Intended Treatment Period": started on day of randomization, ended at efficacy cut-off date (date target number of primary efficacy events [448] was expected to have occurred; set to 30-Jan-2011, prior to unblinding).
Population: Intention to treat analysis, randomized participants. Participants who did not experience an efficacy endpoint event were censored at the earlier of their death date (when death is not part of the endpoint), last contact date (for subjects who withdrew consent to be followed up or were lost to follow-up) or the efficacy cut-off date (30-Jan-2011).
Measure: Number; unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9120 | 9081
participants
  Ischemic or Unspecified Stroke | 159 | 173
  Hemorrhagic Stroke | 38 | 76
  Systemic Embolism | 15 | 16

2. Primary Outcome: Rate of Adjudicated Stroke or Systemic Embolism (SE) During the Intended Treatment Period
Description: Rate=Number of adjudicated stroke or SE events per 100 patient years. Diagnosis of stroke=the nontraumatic focal neurological deficit lasting at least 24 hours, and includes ischemic stroke, hemorrhagic stroke, ischemic stroke with hemorrhagic conversion, stroke of uncertain type, and retinal ischemic event (embolism, infarction). Diagnosis of SE=clinical history consistent with an acute loss of blood flow to a peripheral artery (or arteries), supported by evidence of embolism from surgical specimens, autopsy, angiography, vascular imaging, or other objective testing.
Time Frame: "Intended Treatment Period" started on the day of randomization and ended at the efficacy cut-off date (date on which it was expected that the target number of primary efficacy events [448] would have occurred; set to 30-Jan-2011, prior to unblinding).
Population: as for outcome 1
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9120 | 9081
Number of events per 100 patient years | 1.27 | 1.60
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; With 448 subjects with confirmed strokes or systemic emboli, study would have at least 90% power to meet both regulatory definitions of non-inferiority described in the following: (1) the non-inferiority (NI) of apixaban relative to warfarin was demonstrated if the upper bound of the two-sided 95% confidence interval (CI) for relative risk (RR) was less than 1.38; (2) the NI of apixaban relative to warfarin was demonstrated if the upper bound of the two-sided 99% CI for RR was less than 1.44; Test type: Superiority — With an average 2.1 years follow-up and assuming a stroke rate of 1.20 per hundred patient-years, ~18,000 randomized subjects allocated in a 1:1 ratio to apixaban or warfarin group would be needed to achieve the desired power. These calculations assumed an incidence of 1% loss to follow-up. Non-inferiority for the primary efficacy endpoint will be assessed first. If non-inferiority (using a NI margin of 1.38) is demonstrated then, superiority for the primary efficacy endpoint will be tested; p = 0.0114, Cox Proportional Hazards Model — 2-sided P-value for superiority test; Model included treatment group as a covariate; stratified by investigative site and prior warfarin/vitamin K antagonist status. (experienced, naïve); Hazard Ratio (HR) = 0.79, 95% CI 2-sided [.66 to .95] — apixaban / warfarin

3. Secondary Outcome: Number of Participants With Event of Major (International Society on Thrombosis and Hemostasis [ISTH]) Bleeding During Treatment Period
Description: ISTH Bleeding Criteria: Major bleeding=a bleeding event that was: clinically overt bleeding accompanied by a decrease in hemoglobin (Hgb) of 2 g/dL or more, and/or a transfusion of 2 or more units of packed red blood cells; bleeding that occurred in at least 1 of the following critical sites: intracranial, intraspinal, intraocular (within the corpus of the eye; a conjunctival bleed is not an intraocular bleed), pericardial, intra-articular, intramuscular with compartment syndrome, and retroperitoneal; bleeding that was fatal.
Time Frame: "Treatment Period" started with first dose of blinded study drug and ended 2 days after the last dose of blinded study drug. Mean duration of exposure to double-blind study drug was 1.7 years in each treatment group.
Population: Treated participants. Participants who did not experience a bleeding endpoint were censored at the earlier of 2 days after discontinuation of study drug, or death date, or last-contact date (for participants who withdrew consent to be followed up or were lost to follow-up) at the end of the study.
Measure: Number; unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
participants | 327 | 462

4. Secondary Outcome: Rate of Adjudicated Major (ISTH) Bleed Events During Treatment Period
Description: Rate=number of adjudicated major (ISTH) bleed events per 100 patient years. ISTH Bleeding Criteria: Major bleeding=a bleeding event that was: clinically overt bleeding accompanied by a decrease in hemoglobin (Hgb) of 2 g/dL or more and/or a transfusion of 2 or more units of packed red blood cells; bleeding that occurred in at least 1 of the following sites: intracranial, intraspinal, intraocular (within the corpus of the eye; a conjunctival bleed is not an intraocular bleed), pericardial, intra-articular, intramuscular with compartment syndrome, and retroperitoneal; bleeding that was fatal.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
Number of events per 100 patient years | 2.13 | 3.09
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Test type: Superiority — 4 key objectives were tested using a closed testing procedure. NI for the primary efficacy will be tested 1st. If NI is demonstrated then 1. superiority for the primary efficacy will be tested 2. if superiority for the primary efficacy is 1. not demonstrated, stop 2. demonstrated, then superiority for MB will be tested 3. if superiority for MB is 1. not demonstrated, stop 2. demonstrated, then superiority for all cause death will be tested All tests will be done at 1-sided α = 0.025; p < .0001, Cox Proportional Hazards Model; Model included treatment group as a covariate; stratified by investigative site and prior warfarin/vitamin K antagonist status; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.60 to 0.80] — apixaban / warfarin

5. Secondary Outcome: Number of Participants With Events of All-Cause Death During the Intended Treatment Period
Description: Death was defined as all-cause mortality. All unobserved deaths were assumed to be cardiovascular in nature unless a non-cardiovascular cause could be clearly provided. Cardiovascular=deaths due to ischemic and hemorrhagic stroke, SE, myocardial infarction (MI), sudden death, heart failure, other cardiovascular, and unobserved deaths. Non-cardiovascular=all deaths due to a clearly documented non-cardiovascular cause (further classified into the categories: bleeding, study drug toxicity other than bleeding, malignancy, infection, trauma, and pulmonary causes of death).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9120 | 9081
participants | 603 | 669

6. Secondary Outcome: Rate of Adjudicated All-Cause Death During the Intended Treatment Period
Description: All unobserved deaths were assumed to be cardiovascular in nature unless a non-cardiovascular cause could be clearly provided. Cardiovascular=deaths due to ischemic and hemorrhagic stroke, SE, MI, sudden death, heart failure, other cardiovascular, and unobserved deaths. Non-cardiovascular=all deaths due to a clearly documented non-cardiovascular cause (further classified into the categories: bleeding, study drug toxicity other than bleeding, malignancy, infection, trauma, and pulmonary causes of death).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9120 | 9081
Number of events per 100 patient years | 3.52 | 3.94
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; 4 key objectives were tested using a closed testing procedure. NI for the primary efficacy will be tested 1st. If NI is demonstrated then 1. superiority for the primary efficacy will be tested 2. if superiority for the primary efficacy is 1. not demonstrated, stop 2. demonstrated, then superiority for MB will be tested 3. if superiority for MB is 1. not demonstrated, stop 2. demonstrated, then superiority for all cause death will be tested All tests will be done at 1-sided α = 0.025; Test type: Superiority; p = 0.0465, Cox Proportional Hazards Model; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.80 to 1.00] — apixaban / warfarin

7. Secondary Outcome: Rate of Ischemic or Unspecified Stroke, Hemorrhagic Stroke, Systemic Embolism (SE), and Myocardial Infarction (MI) (as Individual Endpoints) During the Intended Treatment Period
Description: Diagnosis for an acute or evolving MI=elevation of creatine kinase-MB isoenzyme (CK-MB) or Troponin T or I ≥ 2 × the upper limit of normal (ULN), or if no CK-MB or troponin values are available, a total CK ≥ 2×ULN, or new, significant (≥0.04 s) Q waves in ≥2 contiguous leads. For descriptions of Stroke and SE, see Outcome Measure 1.
Time Frame: as for outcome 2
Population: Intention to treat analysis, randomized participants. Participants who did not experience an efficacy endpoint event were censored at the earlier of their death date (when death is not part of the endpoint), last contact date, or the efficacy cut-off date (30-Jan-2011). n=number of participants experiencing stated event.
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9120 | 9081
Number of events per 100 patient years
  Ischemic or Unspecified Stroke (n=162, 175) | 0.97 | 1.05
  Hemorrhagic Stroke (n=40, 78) | 0.24 | 0.47
  Systemic Embolism (n=15, 17) | 0.09 | 0.10
  Myocardial Infarction (n=90, 102) | 0.53 | 0.61
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Ischemic or Unspecified Stroke; Test type: Other; p = 0.4220, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.74 to 1.13] — apixaban / warfarin
Statistical Analysis 2: Comparison: Apixaban vs Warfarin; Hemorrhagic Stroke; Test type: Other; p = 0.0006, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.35 to 0.75] — apixaban / warfarin
Statistical Analysis 3: Comparison: Apixaban vs Warfarin; Systemic Embolism; Test type: Other; p = 0.7020, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.44 to 1.75] — apixaban / warfarin
Statistical Analysis 4: Comparison: Apixaban vs Warfarin; Myocardial Infarction; Test type: Other; p = 0.3720, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.66 to 1.17] — apixaban / warfarin

8. Secondary Outcome: Rate of Ischemic or Unspecified Stroke, Hemorrhagic Stroke, Systemic Embolism (SE), Myocardial Infarction (MI) and All-Cause Death (ACD) (as Composite Endpoints) During the Intended Treatment Period
Description: Diagnosis for an acute or evolving MI=elevation of CK-MB or Troponin T or I ≥ 2 × the ULN, or if no CK-MB or troponin values are available, a total CK ≥ 2×ULN, or new, significant (≥0.04 s) Q waves in ≥2 contiguous leads. For descriptions of Stroke and SE, see Outcome Measure 1. For description of ACD, see Outcome Measure 5.
Time Frame: as for outcome 2
Population: Intention to treat analysis, randomized participants. Participants who didn't experience an efficacy endpoint event were censored at the earlier of their death date (when death is not part of the endpoint), last contact date, or the efficacy cut-off date (30-Jan-2011). n= number of participants experiencing stated combination of events.
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9120 | 9081
Number of events per 100 patient years
  Stroke / SE / Major Bleeding (n=521, 666) | 3.17 | 4.11
  Stroke / SE / All-Cause Death (ACD) (n=752, 837) | 4.49 | 5.04
  Stroke / SE / Major Bleeding / ACD (n=1009, 1168) | 6.13 | 7.20
  Stroke / SE / MI / ACD (n=810, 906) | 4.85 | 5.49
  Ischemic or Unspecified Stroke / ACD (n=725, 796) | 4.32 | 4.78
  Hemorrhagic Stroke / ACD (n=622, 703) | 3.68 | 4.20
  SE / ACD (n=613, 679) | 3.63 | 4.05
  MI / ACD (n=663, 740) | 3.93 | 4.43
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Composite of Stroke / Systemic Embolism / Major Bleeding; Test type: Other; p < .0001, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.69 to 0.86] — apixaban / warfarin
Statistical Analysis 2: Comparison: Apixaban vs Warfarin; Composite of Stroke / Systemic Embolism / All-Cause Death; Test type: Other; p = 0.0192, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.81 to 0.98] — apixaban / warfarin
Statistical Analysis 3: Comparison: Apixaban vs Warfarin; Composite of Stroke / Systemic Embolism / Major Bleeding / All-Cause Death; Test type: Other; p = 0.0002, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.78 to 0.92] — apixaban / warfarin
Statistical Analysis 4: Comparison: Apixaban vs Warfarin; Composite of Stroke / Systemic Embolism / MI / All-Cause Death; Test type: Other; p = 0.0107, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.80 to 0.97] — apixaban / warfarin
Statistical Analysis 5: Comparison: Apixaban vs Warfarin; Composite of Ischemic or Unspecified Stroke / All-Cause Death; Test type: Other; p = 0.0432, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.82 to 1.00] — apixaban / warfarin
Statistical Analysis 6: Comparison: Apixaban vs Warfarin; Composite of Hemorrhagic Stroke / All-Cause Death; Test type: Other; p = 0.0167, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.79 to 0.98] — apixaban / warfarin
Statistical Analysis 7: Comparison: Apixaban vs Warfarin; Composite of Systemic Embolism / All-Cause Death; Test type: Other; p = 0.0464, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.80 to 1.00] — apixaban / warfarin
Statistical Analysis 8: Comparison: Apixaban vs Warfarin; Composite of Myocardial Infarction / All-Cause Death; Test type: Other; p = 0.0253, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.80 to 0.99] — apixaban / warfarin

9. Secondary Outcome: Number of Warfarin/Vitamin K Antagonist (VKA) Naive Participants With Composite Stroke / Systemic Embolism (SE) / Major Bleeding During the Intended Treatment Period
Description: For descriptions of Stroke and SE, see Outcome Measure 1. For description of Major bleeding, see Outcome Measure 3.
Time Frame: as for outcome 2
Population: Intention to treat analysis, randomized participants who were Warfarin/Vitamin K Antagonist (VKA) naïve (a stratification variable, defined as receiving ≤30 consecutive days of prior warfarin/VKA treatment). Participants not experiencing efficacy endpoint event were censored at earlier of death, last contact, or efficacy cut-off date (30-Jan-2011).
Measure: Number; unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 3912 | 3888
participants | 229 | 285

10. Secondary Outcome: Rate of Composite Stroke / Systemic Embolism / Major Bleeding in Warfarin/Vitamin K Antagonist (VKA) Naive Participants During the Intended Treatment Period
Time Frame: as for outcome 2
Population: Intention to treat analysis, randomized participants. Participants who did not experience an efficacy endpoint event were censored at the earlier of their death date, last contact date, or the efficacy cut-off date (30-Jan-2011).
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 3912 | 3888
Number of events per 100 patient years | 3.21 | 4.06
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Composite Stroke/Systemic Embolism/Major Bleeding in Warfarin/Vitamin K Antagonist (VKA) Naive Participants; Test type: Other; p = 0.0098, Cox Proportional Hazards Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.67 to 0.95] — apixaban / warfarin

11. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs), Bleeding AEs, Serious Adverse Events (SAEs), Discontinuations Due to AEs, or Deaths During the Treatment Period
Description: AE: all SAEs or AEs with onset from first dose through 2 days (AEs) or 30 days (SAEs) after the last dose of blinded study drug (BSD). SAE: all SAEs with onset from first dose through 30 days after the last dose of BSD. Bleeding AE: all serious or non-serious bleeding-related AEs with onset from first dose through 2 days after the last dose of BSD. Discontinuations due to AE: all SAEs or AEs with onset from first dose of BSD and with action taken=drug discontinued. Deaths: all deaths occurring from first dose through 30 days after the last dose of BSD.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
participants
  AE | 7406 | 7521
  SAE | 3182 | 3302
  Bleeding AE | 2288 | 2961
  Discontinuations due to AE | 688 | 758
  Deaths | 429 | 468

12. Secondary Outcome: Number of Participants With Events of Major or Clinically Relevant Nonmajor (CRNM) Bleed During Treatment Period
Description: Major bleeding=bleeding that is clinically overt and that either resulted in a decrease in hemoglobin of 2 g/dL or more over a 24-hour period, led to a transfusion of 2 or more units of packed red blood cells, occurred in a critical site, or led to death. CRNM bleeding=bleeding that is clinically overt, that satisfies none of the additional criteria required for the event to be adjudicated as a major bleeding event, that led to either hospital admission for bleeding, physician-guided medical or surgical treatment for bleeding, or a change in antithrombotic therapy.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
participants | 613 | 877

13. Secondary Outcome: Rate of Events of Major or Clinically Relevant Non-Major (CRNM) Bleed During Treatment Period
Description: Rate=number of major or CRNM bleed events per 100 patient years. Major=clinically overt and either 1) resulted in a decrease in hemoglobin of 2 g/dL or more, or 2) led to a transfusion of 2 or more units of packed red blood cells, or 3) occurred in a critical site, or 4) led to death. CRNM bleeding=clinically overt, but satisfied no additional criteria required to be adjudicated as a major bleeding event, and led to either 1) hospital admission for bleeding or 2) physician guided medical or surgical treatment for bleeding or 3) a change in antithrombotic therapy.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: number of events / 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
number of events / 100 patient years | 4.07 | 6.01
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Test type: Other; p < .0001, Cox Proportional Hazard Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.61 to 0.75] — apixaban / warfarin

14. Secondary Outcome: Number of Participants With All Bleeding Events During Treatment Period
Description: All bleeding events include major bleeding, CRNM bleeding (see Outcome Measure 12 Description for definitions), plus events of minor bleeding and fatal bleeding. Minor bleeding: All acute clinically overt bleeding events not meeting the criteria for either major bleeding or clinically relevant non-major bleeding will be classified as minor bleeding. Fatal bleeding is defined as a bleeding event that the Clinical Events Committee determines is the primary cause of death or contributes directly to death.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
participants | 2356 | 3060

15. Secondary Outcome: Rate of All Bleeding Events During Treatment Period
Description: Rate=number of all bleeding events per 100 patient years. "All bleeding events" include major bleeding, CRNM bleeding (see Outcome Measure 12 Description for definitions), plus events of minor bleeding and fatal bleeding. Minor bleeding: All acute clinically overt bleeding events not meeting the criteria for either major bleeding or clinically relevant non-major bleeding will be classified as minor bleeding. Fatal bleeding is defined as a bleeding event that the Clinical Events Committee determines is the primary cause of death or contributes directly to death.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
number of events per 100 patient years | 18.08 | 25.82
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Test type: Other; p < .0001, Cox Proportional Hazard Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.68 to 0.75] — apixaban / warfarin

16. Other Pre Specified Outcome: Rate of Adjudicated Bleeding Endpoints Per Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) During the Treatment Period
Description: Rate=number of adjudicated GUSTO bleeding events per 100 patient years. GUSTO Bleeding Criteria: GUSTO severe (or life-threatening) bleeding: either intracranial hemorrhage or bleeding that causes hemodynamic compromise and requires intervention. GUSTO moderate bleeding: bleeding that requires blood transfusion but does not result in hemodynamic compromise.
Time Frame: as for outcome 3
Population: Treated participants. Participants who did not experience a bleeding endpoint were censored at the earlier of 2 days after discontinuation of study drug, or death date, or last-contact date (for participants who withdrew consent to be followed up or were lost to follow-up) at the end of the study. n=number of participants experiencing events.
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
Number of events per 100 patient years
  Severe (n=80, 172)) | 0.52 | 1.13
  Severe or Moderate (n=199, 328) | 1.29 | 2.18
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Severe GUSTO bleeding events; Test type: Other; p < .0001, Cox Proportional Hazard Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.35 to 0.60] — apixaban / warfarin
Statistical Analysis 2: Comparison: Apixaban vs Warfarin; Severe or Moderate GUSTO bleeding events; Test type: Other; p < .0001, Cox Proportional Hazard Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.50 to 0.71] — apixaban / warfarin

17. Other Pre Specified Outcome: Rate of Adjudicated Bleeding Endpoints Per Thrombolysis in Myocardial Infarction (TIMI) During the Treatment Period
Description: Rate=number of adjudicated TIMI bleeding events per 100 patient years. TIMI Bleeding Criteria: Major bleeding=Intracranial bleeding and/or clinically overt bleeding associated with ≥5 gm/dL fall in Hgb or 15% fall in hematocrit (Hct) from baseline, accounting for transfusions. Minor bleeding=Clinically overt bleeding associated with ≥3 gm/dL fall in Hgb or a ≥10% fall in Hct from baseline, accounting for transfusions.
Time Frame: as for outcome 3
Population: as for outcome 16
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
Number of events per 100 patient years
  Major (n=148, 256) | 0.96 | 1.69
  Major or Minor (n=239, 370) | 1.55 | 2.46
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Major TIMI bleeding event; Test type: Other; p < .0001, Cox Proportional Hazard Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.46 to 0.70] — apixaban / warfarin
Statistical Analysis 2: Comparison: Apixaban vs Warfarin; Major or Minor TIMI bleeding criteria; Test type: Other; p < .0001, Cox Proportional Hazard Model; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.54 to 0.75] — apixaban / warfarin

18. Other Pre Specified Outcome: Number of Participants With Net-Clinical Benefit During Treatment Period
Description: Net-Clinical Benefit = Composite of stroke, systemic embolism and ISTH major bleeding.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
participants | 459 | 608

19. Other Pre Specified Outcome: Rate of Net-Clinical Benefit During Treatment Period
Description: Rate=number of events of net-clinical benefit per 100 patient years. Net-Clinical Benefit = Composite of stroke, systemic embolism and ISTH major bleeding
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number; unit: Number of events per 100 patient years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 9088 | 9052
Number of events per 100 patient years | 3.01 | 4.09
Statistical Analysis 1: Comparison: Apixaban vs Warfarin; Test type: Other; p < .0001, Cox Proportional Hazard Model — nominal two-sided p-value was associated with a test of H0: RR=1 vs H1: RR ≠ 1; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.65 to 0.83] — apixaban / warfarin

ADVERSE EVENTS:
Description: Treated population (includes all patients who received at least 1 dose of study drug.)
Arm/Group | Warfarin | Apixaban
Serious Adverse Events (participants affected / at risk) | 3182/9088 | 3302/9052
Other Adverse Events (participants affected / at risk) | 3876/9088 | 4071/9052
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin (N=9088) | Apixaban (N=9052)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 2
Abscess limb (Infections and infestations) | 3 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 4
Acid fast bacilli infection (Infections and infestations) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 20 | 16
Acute megakaryocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Alcohol abuse (Psychiatric disorders) | 4 | 2
Anxiety disorder (Psychiatric disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 7 | 6
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Atrial fibrillation (Cardiac disorders) | 301 | 287
Balance disorder (Nervous system disorders) | 0 | 1
Balanitis (Reproductive system and breast disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Cardiac fibrillation (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 6 | 4
Carotid arteriosclerosis (Nervous system disorders) | 2 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Cataract nuclear (Eye disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 3
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 15 | 18
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 5 | 3
Circulatory collapse (Vascular disorders) | 3 | 4
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cor pulmonale (Cardiac disorders) | 2 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 1
Device battery issue (General disorders) | 2 | 3
Device failure (General disorders) | 3 | 2
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Drug interaction (General disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 6
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 3 | 3
Endocarditis (Infections and infestations) | 0 | 2
Epilepsy (Nervous system disorders) | 7 | 6
Femoral artery embolism (Vascular disorders) | 1 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Gangrene (Infections and infestations) | 5 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 11
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 9 | 10
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Haematemesis (Gastrointestinal disorders) | 1 | 4
Haematuria (Renal and urinary disorders) | 34 | 44
Haemodynamic instability (Vascular disorders) | 1 | 1
Haemoglobin decreased (Investigations) | 3 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1
Haemorrhoid infection (Infections and infestations) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 2
Heart rate increased (Investigations) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Herpes zoster infection neurological (Infections and infestations) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 2
Hypertensive encephalopathy (Nervous system disorders) | 0 | 2
Hypotonia (Nervous system disorders) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 3 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 3
Implant site inflammation (General disorders) | 0 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Incision site infection (Infections and infestations) | 1 | 2
Infected epidermal cyst (Infections and infestations) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 20 | 29
Intercostal neuralgia (Nervous system disorders) | 1 | 0
International normalised ratio increased (Investigations) | 3 | 5
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral discitis (Infections and infestations) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 8 | 1
Large intestinal ulcer (Gastrointestinal disorders) | 0 | 2
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Left ventricular failure (Cardiac disorders) | 7 | 9
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 2
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lobar pneumonia (Infections and infestations) | 16 | 12
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 12 | 12
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 2
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0
Occult blood (Investigations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 2
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 4 | 4
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 3 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 2
Peripheral artery aneurysm (Vascular disorders) | 1 | 1
Peripheral vascular disorder (Vascular disorders) | 3 | 5
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Phacolytic glaucoma (Eye disorders) | 1 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonia (Infections and infestations) | 202 | 231
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound infection (Infections and infestations) | 3 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 1
Prostatic specific antigen increased (Investigations) | 0 | 2
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 1 | 0
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 | 1
Retinal vascular occlusion (Eye disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 | 4
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 3
Sinus bradycardia (Cardiac disorders) | 6 | 3
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 4
Splenic injury (Injury, poisoning and procedural complications) | 0 | 1
Staphylococcal infection (Infections and infestations) | 3 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Subdiaphragmatic abscess (Infections and infestations) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 13 | 14
Treatment noncompliance (Social circumstances) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Typhoid fever (Infections and infestations) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 23 | 32
Upper limb fracture (Injury, poisoning and procedural complications) | 6 | 7
Uraemic encephalopathy (Nervous system disorders) | 1 | 0
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 3
Adrenal haemorrhage (Endocrine disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 1
Aneurysm ruptured (Vascular disorders) | 0 | 1
Angiodysplasia (Vascular disorders) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 3 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 3
Blood glucose abnormal (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Bloody discharge (General disorders) | 0 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cellulitis (Infections and infestations) | 1 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchopneumonia (Infections and infestations) | 9 | 7
Bundle branch block left (Cardiac disorders) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 4
Carotid sinus syndrome (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 20 | 27
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 19 | 19
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 3 | 5
Colitis ischaemic (Gastrointestinal disorders) | 3 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 5
Cystitis noninfective (Renal and urinary disorders) | 0 | 2
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Device dislocation (General disorders) | 2 | 4
Device related infection (Infections and infestations) | 6 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 19 | 28
Diabetic microangiopathy (Vascular disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 2
Dizziness postural (Nervous system disorders) | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Empyema (Infections and infestations) | 2 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Endometritis (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 4 | 4
Foot fracture (Injury, poisoning and procedural complications) | 4 | 0
Gastritis (Gastrointestinal disorders) | 17 | 8
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 2 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Glaucoma (Eye disorders) | 0 | 6
Gout (Metabolism and nutrition disorders) | 11 | 9
Grand mal convulsion (Nervous system disorders) | 2 | 1
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 9 | 11
Hallucination, visual (Psychiatric disorders) | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hepatic enzyme increased (Investigations) | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 2
Hypocoagulable state (Blood and lymphatic system disorders) | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1
Iliac artery stenosis (Vascular disorders) | 0 | 2
Implant site infection (Infections and infestations) | 1 | 0
Intermittent claudication (Vascular disorders) | 4 | 3
Intestinal obstruction (Gastrointestinal disorders) | 3 | 9
Intracardiac thrombus (Cardiac disorders) | 2 | 1
Klebsiella test positive (Investigations) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 4 | 1
Lip haemorrhage (Gastrointestinal disorders) | 1 | 2
Liver abscess (Infections and infestations) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 1
Malaria (Infections and infestations) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 2
Mastitis (Infections and infestations) | 0 | 1
Medical device site reaction (General disorders) | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 80 | 63
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 22 | 26
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oedema (General disorders) | 2 | 1
Oesophageal disorder (Gastrointestinal disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 4 | 10
Otitis media (Infections and infestations) | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 8 | 4
Panic attack (Psychiatric disorders) | 1 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 2
Periodontitis (Gastrointestinal disorders) | 2 | 1
Peripheral embolism (Vascular disorders) | 6 | 4
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 2 | 2
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyp colorectal (Gastrointestinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 9 | 5
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Respiratory tract infection (Infections and infestations) | 17 | 16
Retinal vein thrombosis (Eye disorders) | 4 | 0
Schamberg's disease (Skin and subcutaneous tissue disorders) | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 2
Sinus arrest (Cardiac disorders) | 4 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 4 | 8
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Staphylococcus test positive (Investigations) | 1 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 5
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Thrombosis (Vascular disorders) | 0 | 4
Tooth socket haemorrhage (Gastrointestinal disorders) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 2
Traumatic arthropathy (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 3 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 2
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 2
VIIth nerve paralysis (Nervous system disorders) | 2 | 2
Varicose vein ruptured (Vascular disorders) | 1 | 0
Vesical fistula (Renal and urinary disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 1
Weight increased (Investigations) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 1
Adrenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal prolapse (Gastrointestinal disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 112 | 87
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 2 | 2
Arterial restenosis (Injury, poisoning and procedural complications) | 1 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Asherman's syndrome (Reproductive system and breast disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Ataxia (Nervous system disorders) | 2 | 3
Atrial thrombosis (Cardiac disorders) | 4 | 2
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Bile duct stone (Hepatobiliary disorders) | 4 | 5
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 13
Bladder mass (Renal and urinary disorders) | 0 | 1
Bladder neck obstruction (Renal and urinary disorders) | 3 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Blood pressure increased (Investigations) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bradyarrhythmia (Cardiac disorders) | 9 | 3
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchitis haemophilus (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 1
Cardiac valve disease (Cardiac disorders) | 2 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 3
Chest discomfort (General disorders) | 4 | 2
Chronic hepatitis (Hepatobiliary disorders) | 1 | 0
Coagulation time prolonged (Investigations) | 6 | 9
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 26
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Cyanosis (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 11 | 14
Dehydration (Metabolism and nutrition disorders) | 25 | 27
Dementia Alzheimer's type (Nervous system disorders) | 0 | 4
Dental caries (Gastrointestinal disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 8
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 4 | 2
Endocarditis bacterial (Infections and infestations) | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 2
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Erysipelas (Infections and infestations) | 12 | 15
Extrasystoles (Cardiac disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 4 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 24 | 30
Fibrosis (General disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 13 | 12
Gastritis erosive (Gastrointestinal disorders) | 5 | 9
Gastritis haemorrhagic (Gastrointestinal disorders) | 5 | 7
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Hepatic congestion (Hepatobiliary disorders) | 2 | 2
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 2 | 2
Hernia (General disorders) | 2 | 1
Hypertensive crisis (Vascular disorders) | 16 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 15 | 8
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Implant site reaction (General disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Injection site abscess (Infections and infestations) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 3 | 2
Intestinal polyp (Gastrointestinal disorders) | 1 | 3
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 1
Jejunal perforation (Gastrointestinal disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Laryngitis (Infections and infestations) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 4 | 4
Leriche syndrome (Vascular disorders) | 1 | 0
Liver function test abnormal (Investigations) | 6 | 2
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Lymphoedema (Vascular disorders) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 3
Mitral valve disease (Cardiac disorders) | 1 | 1
Multi-organ failure (General disorders) | 5 | 5
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 3 | 0
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Necrosis ischaemic (Vascular disorders) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Open fracture (Injury, poisoning and procedural complications) | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 11 | 13
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 2 | 2
Phimosis (Congenital, familial and genetic disorders) | 1 | 4
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Prostate examination abnormal (Investigations) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Psychosomatic disease (Psychiatric disorders) | 1 | 0
Radiculitis cervical (Nervous system disorders) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 11
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal arteriosclerosis (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5 | 4
Right ventricular failure (Cardiac disorders) | 5 | 2
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal cord ischaemia (Nervous system disorders) | 0 | 1
Spinal vascular disorder (Nervous system disorders) | 0 | 1
Splenic cyst (Blood and lymphatic system disorders) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 2
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 2
Sudden death (General disorders) | 57 | 50
Syringomyelia (Nervous system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 7
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 5 | 3
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 1
Tuberculosis (Infections and infestations) | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 11
Urethritis (Infections and infestations) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 2
Ventricular arrhythmia (Cardiac disorders) | 2 | 4
Ventricular fibrillation (Cardiac disorders) | 9 | 12
Vertigo positional (Ear and labyrinth disorders) | 1 | 4
Weight decreased (Investigations) | 0 | 3
Weil's disease (Infections and infestations) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal wall disorder (Gastrointestinal disorders) | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adverse drug reaction (General disorders) | 2 | 1
Amaurosis (Eye disorders) | 0 | 1
Amyloidosis (Immune system disorders) | 1 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angina pectoris (Cardiac disorders) | 49 | 39
Ankle fracture (Injury, poisoning and procedural complications) | 9 | 9
Aortic dissection (Vascular disorders) | 1 | 3
Aortic valve stenosis (Cardiac disorders) | 7 | 1
Appendicitis (Infections and infestations) | 13 | 9
Arterial haemorrhage (Vascular disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 9 | 6
Ascites (Gastrointestinal disorders) | 3 | 2
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Atrioventricular block (Cardiac disorders) | 5 | 3
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Bacterial infection (Infections and infestations) | 0 | 1
Basedow's disease (Endocrine disorders) | 1 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 26 | 24
Biliary colic (Hepatobiliary disorders) | 3 | 2
Bleeding varicose vein (Vascular disorders) | 1 | 0
Blood amylase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood osmolarity decreased (Investigations) | 1 | 0
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Cardiac disorder (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 8 | 8
Cardiogenic shock (Cardiac disorders) | 9 | 7
Cerebrosclerosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 35 | 51
Cerebrovascular disorder (Nervous system disorders) | 4 | 9
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 2
Chest injury (Injury, poisoning and procedural complications) | 1 | 3
Cholecystitis acute (Hepatobiliary disorders) | 16 | 20
Cholestasis (Hepatobiliary disorders) | 1 | 1
Chronic lymphocytic leukaemia stage 2 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 5
Coagulation test abnormal (Investigations) | 1 | 0
Coronary artery dissection (Cardiac disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Critical illness polyneuropathy (Nervous system disorders) | 0 | 1
Cystitis (Infections and infestations) | 3 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Device malfunction (General disorders) | 11 | 6
Diabetic coma (Nervous system disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 1
Dysentery (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Embolism (Vascular disorders) | 4 | 3
Embolism arterial (Vascular disorders) | 1 | 0
Encephalitis (Nervous system disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 3
Eyelid ptosis (Eye disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 9 | 4
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 2
Gallstone ileus (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 5 | 6
Gastroenteritis viral (Infections and infestations) | 3 | 5
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
H1N1 influenza (Infections and infestations) | 2 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 3 | 6
Haematochezia (Gastrointestinal disorders) | 4 | 7
Haemoglobin abnormal (Investigations) | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 6 | 9
Hepatitis toxic (Hepatobiliary disorders) | 1 | 1
Hernia obstructive (General disorders) | 3 | 2
Hydrocephalus (Nervous system disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 9
Hyperthyroidism (Endocrine disorders) | 3 | 4
Hypertonia (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Ileus (Gastrointestinal disorders) | 4 | 5
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 2
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Infected bites (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
International normalised ratio fluctuation (Investigations) | 0 | 1
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 5 | 6
Joint sprain (Injury, poisoning and procedural complications) | 2 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipase increased (Investigations) | 0 | 2
Localised infection (Infections and infestations) | 2 | 3
Lower respiratory tract infection (Infections and infestations) | 20 | 10
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung infection (Infections and infestations) | 8 | 11
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 23
Lymphorrhoea (Vascular disorders) | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8
Malnutrition (Metabolism and nutrition disorders) | 0 | 2
Mass (General disorders) | 3 | 0
Mastoiditis (Infections and infestations) | 0 | 1
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 10 | 8
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 17 | 17
Necrobiosis (General disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 5 | 8
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 26 | 40
Pallor (Vascular disorders) | 0 | 1
Paranoia (Psychiatric disorders) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 4 | 2
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 1 | 1
Peritoneal infection (Infections and infestations) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Podagra (Metabolism and nutrition disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 3 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostatic dysplasia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 2 | 3
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pyelonephritis (Infections and infestations) | 8 | 1
Renal failure acute (Renal and urinary disorders) | 57 | 35
Renal impairment (Renal and urinary disorders) | 3 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 26 | 22
Skull fracture (Injury, poisoning and procedural complications) | 0 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 23
Subdural haematoma (Injury, poisoning and procedural complications) | 7 | 27
Suicidal ideation (Psychiatric disorders) | 0 | 1
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 2
Tooth abscess (Infections and infestations) | 3 | 3
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Umbilical hernia (Gastrointestinal disorders) | 1 | 8
Urinary retention (Renal and urinary disorders) | 11 | 7
Vascular rupture (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 3
Vertebrobasilar insufficiency (Nervous system disorders) | 7 | 7
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1
Vitreous degeneration (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 3 | 4
Wrist fracture (Injury, poisoning and procedural complications) | 4 | 2
Abscess (Infections and infestations) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 11 | 15
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 48 | 43
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 2
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 1
Anal fistula infection (Infections and infestations) | 0 | 1
Anal skin tags (Gastrointestinal disorders) | 0 | 1
Angiopathy (Vascular disorders) | 1 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 4 | 0
Arterial thrombosis (Vascular disorders) | 1 | 3
Arthritis bacterial (Infections and infestations) | 6 | 3
Arthritis infective (Infections and infestations) | 4 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Barotrauma (Injury, poisoning and procedural complications) | 1 | 0
Basilar artery thrombosis (Nervous system disorders) | 1 | 0
Bladder stenosis (Renal and urinary disorders) | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 1
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Breast calcifications (Reproductive system and breast disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 19
Breast hyperplasia (Reproductive system and breast disorders) | 1 | 0
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 3 | 2
Calculus urinary (Renal and urinary disorders) | 6 | 6
Cardiac amyloidosis (Cardiac disorders) | 0 | 1
Cardiac death (General disorders) | 11 | 6
Cardiac failure chronic (Cardiac disorders) | 16 | 23
Cardiac failure congestive (Cardiac disorders) | 171 | 175
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 6 | 7
Cataract (Eye disorders) | 26 | 34
Cellulitis (Infections and infestations) | 44 | 60
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 3
Cholangitis (Hepatobiliary disorders) | 5 | 4
Cholecystitis infective (Infections and infestations) | 3 | 3
Coagulopathy (Blood and lymphatic system disorders) | 4 | 6
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Coma (Nervous system disorders) | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 8 | 8
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Cutis laxa (Skin and subcutaneous tissue disorders) | 0 | 1
Death (General disorders) | 16 | 26
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Device lead damage (General disorders) | 3 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 1 | 1
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 1
Diverticulum (Gastrointestinal disorders) | 5 | 5
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 6
Drug administration error (Injury, poisoning and procedural complications) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Endocarditis haemophilus (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 2 | 0
Escherichia bacteraemia (Infections and infestations) | 2 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 0
Eyeball rupture (Injury, poisoning and procedural complications) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 11 | 16
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gait disturbance (General disorders) | 1 | 2
Gastroenteritis (Infections and infestations) | 30 | 21
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 3
HIV test positive (Investigations) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 21
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 5 | 3
Haemorrhagic stroke (Nervous system disorders) | 22 | 40
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 3 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Headache (Nervous system disorders) | 5 | 1
Heart valve stenosis (Cardiac disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 3
Hernial eventration (Gastrointestinal disorders) | 0 | 2
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 19 | 28
Homicide (Social circumstances) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 5 | 2
Hyperaldosteronism (Endocrine disorders) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 2
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 18 | 14
Impaired healing (General disorders) | 0 | 1
Implant site thrombosis (General disorders) | 0 | 1
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 3 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 2
Intracranial haematoma (Nervous system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 | 9
Ischaemia (Vascular disorders) | 1 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 2
Ischaemic ulcer (General disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 3 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 2 | 0
Lacunar infarction (Nervous system disorders) | 6 | 4
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Localised oedema (General disorders) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 4
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Medical device complication (General disorders) | 2 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Neurilemmoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 1
Ocular vascular disorder (Eye disorders) | 1 | 0
Oedema peripheral (General disorders) | 6 | 5
Open angle glaucoma (Eye disorders) | 0 | 2
Oral infection (Infections and infestations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 69 | 63
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Panic disorder (Psychiatric disorders) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 4 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Perineal abscess (Infections and infestations) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 15
Pilonidal cyst (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Primary hyperaldosteronism (Endocrine disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 | 35
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Prostatism (Reproductive system and breast disorders) | 4 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Pyelonephritis acute (Infections and infestations) | 3 | 3
Pyelonephritis chronic (Infections and infestations) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 19 | 19
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal colic (Renal and urinary disorders) | 4 | 4
Renal failure (Renal and urinary disorders) | 23 | 22
Retinal artery occlusion (Eye disorders) | 2 | 2
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salmonellosis (Infections and infestations) | 1 | 0
Sensory disturbance (Nervous system disorders) | 1 | 1
Shock (Vascular disorders) | 4 | 5
Spinal claudication (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 2
Streptococcal infection (Infections and infestations) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 6 | 9
Subileus (Gastrointestinal disorders) | 0 | 1
Sudden cardiac death (General disorders) | 30 | 18
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 5
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 3 | 3
Traumatic renal injury (Injury, poisoning and procedural complications) | 2 | 1
Urinary bladder polyp (Renal and urinary disorders) | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Vascular encephalopathy (Nervous system disorders) | 2 | 4
Venous insufficiency (Vascular disorders) | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Wallenberg syndrome (Nervous system disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 14 | 13
Abdominal sepsis (Infections and infestations) | 0 | 2
Acquired oesophageal web (Gastrointestinal disorders) | 0 | 1
Adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Alveolitis fibrosing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Amnesia (Nervous system disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 3 | 0
Aortic rupture (Vascular disorders) | 0 | 2
Aortic stenosis (Vascular disorders) | 12 | 8
Aphakia (Eye disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 12
Arteriosclerosis (Vascular disorders) | 4 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 7 | 12
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30 | 35
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Brain stem infarction (Nervous system disorders) | 0 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bronchitis bacterial (Infections and infestations) | 0 | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 5 | 2
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 9 | 7
Catheterisation cardiac (Investigations) | 2 | 0
Chest pain (General disorders) | 43 | 72
Chorioretinal disorder (Eye disorders) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Chronotropic incompetence (Cardiac disorders) | 0 | 1
Clostridium test positive (Investigations) | 1 | 1
Colitis (Gastrointestinal disorders) | 4 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 2
Conduction disorder (Cardiac disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 9 | 3
Crush syndrome (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Dacryocystitis (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 7 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 4
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Dizziness (Nervous system disorders) | 18 | 13
Drug level increased (Investigations) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 3 | 1
Epididymitis (Reproductive system and breast disorders) | 2 | 1
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Eye disorder (Eye disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Frontotemporal dementia (Nervous system disorders) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 1
Gastroenteritis shigella (Infections and infestations) | 0 | 1
Granuloma (General disorders) | 1 | 1
Haematoma (Vascular disorders) | 16 | 37
Haemorrhage (Vascular disorders) | 7 | 10
Head injury (Injury, poisoning and procedural complications) | 6 | 13
Hemiparesis (Nervous system disorders) | 2 | 2
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Hepatic ischaemia (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 5
Hepatitis B (Infections and infestations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 38 | 30
Hypothyroidism (Endocrine disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Infected skin ulcer (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 5 | 11
Infusion site haemorrhage (General disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Intra-abdominal haematoma (Vascular disorders) | 0 | 1
Intra-abdominal haemorrhage (Vascular disorders) | 1 | 3
Ischaemic stroke (Nervous system disorders) | 91 | 76
Joint abscess (Infections and infestations) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 | 6
Lung abscess (Infections and infestations) | 0 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Macular oedema (Eye disorders) | 0 | 1
Malaise (General disorders) | 3 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Migraine with aura (Nervous system disorders) | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 4 | 4
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Pancoast's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 1
Paralysis (Nervous system disorders) | 1 | 1
Paranasal sinus benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 0
Phlebitis (Vascular disorders) | 2 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1
Postrenal failure (Renal and urinary disorders) | 1 | 1
Presyncope (Nervous system disorders) | 15 | 12
Prostatic disorder (Reproductive system and breast disorders) | 1 | 2
Psychotic disorder (Psychiatric disorders) | 0 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Renal injury (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 2 | 2
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Retinal detachment (Eye disorders) | 5 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 5 | 1
Scrotal swelling (Reproductive system and breast disorders) | 1 | 0
Sedation (Nervous system disorders) | 0 | 1
Septic shock (Infections and infestations) | 5 | 7
Serum sickness (Immune system disorders) | 0 | 1
Sinobronchitis (Infections and infestations) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 2 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Staphylococcal sepsis (Infections and infestations) | 3 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 1
Superinfection (Infections and infestations) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 6 | 4
Surgical procedure repeated (Injury, poisoning and procedural complications) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 60 | 39
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 3
Tricuspid valve incompetence (Cardiac disorders) | 2 | 2
Troponin increased (Investigations) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 1
Ulcer haemorrhage (General disorders) | 1 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 3
Urinary tract infection (Infections and infestations) | 60 | 48
Uterine abscess (Infections and infestations) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Uterine polyp (Reproductive system and breast disorders) | 5 | 0
Varicose vein (Vascular disorders) | 3 | 5
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 5
Venous thrombosis limb (Vascular disorders) | 2 | 2
Ventricular tachycardia (Cardiac disorders) | 27 | 31
Vestibulitis (General disorders) | 1 | 0
Viral infection (Infections and infestations) | 3 | 3
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Wound infection (Infections and infestations) | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 9 | 3
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 3
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 44 | 44
Acute sinusitis (Infections and infestations) | 0 | 1
Adams-Stokes syndrome (Cardiac disorders) | 1 | 1
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 6
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Anticonvulsant drug level below therapeutic (Investigations) | 0 | 1
Anxiety (Psychiatric disorders) | 9 | 1
Aortic valve disease (Cardiac disorders) | 0 | 2
Appendiceal abscess (Infections and infestations) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 2
Arteriosclerosis obliterans (Vascular disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 29 | 35
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder diverticulum (Renal and urinary disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Bradycardia (Cardiac disorders) | 32 | 43
Brain abscess (Infections and infestations) | 1 | 0
Brain injury (Nervous system disorders) | 0 | 1
Brain stem haemorrhage (Nervous system disorders) | 0 | 3
Cardiac asthma (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 310 | 301
Cellulitis of male external genital organ (Infections and infestations) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 4 | 2
Chills (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 24 | 16
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 68 | 76
Clostridial infection (Infections and infestations) | 2 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 11 | 12
Complex partial seizures (Nervous system disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 6 | 4
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery disease (Cardiac disorders) | 60 | 61
Cyst (General disorders) | 0 | 1
Dementia (Nervous system disorders) | 3 | 3
Diabetic neuropathy (Nervous system disorders) | 2 | 3
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diverticulitis (Infections and infestations) | 13 | 12
Drug hypersensitivity (Immune system disorders) | 1 | 1
Dural tear (Injury, poisoning and procedural complications) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 2
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Femoral arterial stenosis (Vascular disorders) | 2 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 2 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Gastrointestinal erosion (Gastrointestinal disorders) | 0 | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 2 | 3
Goitre (Endocrine disorders) | 3 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Haematocrit decreased (Investigations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 2
Heart rate decreased (Investigations) | 0 | 1
Heart valve incompetence (Cardiac disorders) | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 4 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 11 | 5
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 0 | 1
Infected sebaceous cyst (Infections and infestations) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 2 | 3
International normalised ratio abnormal (Investigations) | 5 | 5
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 8 | 10
Intestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 3
Keratitis sclerosing (Eye disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 6
Limb injury (Injury, poisoning and procedural complications) | 2 | 1
Liver disorder (Hepatobiliary disorders) | 2 | 1
Loss of consciousness (Nervous system disorders) | 0 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Migraine (Nervous system disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 13 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Myasthenia gravis (Nervous system disorders) | 0 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Myoglobinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Nerve root lesion (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 1 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nosocomial infection (Infections and infestations) | 0 | 1
Occult blood positive (Investigations) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Organ failure (General disorders) | 0 | 1
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic mass (General disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Pericarditis (Cardiac disorders) | 1 | 3
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 3
Polyp (General disorders) | 2 | 2
Post procedural infection (Infections and infestations) | 0 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 1
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22 | 21
Puncture site haemorrhage (General disorders) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal aneurysm (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 1
Renal embolism (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 4 | 10
Respiratory tract infection viral (Infections and infestations) | 0 | 2
Retinal haemorrhage (Eye disorders) | 3 | 3
Retinopathy (Eye disorders) | 0 | 1
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 7 | 12
Sick sinus syndrome (Cardiac disorders) | 49 | 40
Skin ulcer (Skin and subcutaneous tissue disorders) | 8 | 5
Small intestinal obstruction (Gastrointestinal disorders) | 8 | 13
Spinal haematoma (Nervous system disorders) | 1 | 0
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Syncope (Nervous system disorders) | 79 | 49
Thalassaemia beta (Congenital, familial and genetic disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 5 | 6
Ureteric perforation (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 2 | 4
Urinary tract obstruction (Renal and urinary disorders) | 2 | 1
Urosepsis (Infections and infestations) | 16 | 7
Vascular dementia (Nervous system disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 21 | 13
Victim of homicide (Social circumstances) | 0 | 1
Volvulus (Gastrointestinal disorders) | 2 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 2 | 1
Abdominal abscess (Infections and infestations) | 2 | 2
Abdominal adhesions (Gastrointestinal disorders) | 1 | 2
Abdominal hernia (Gastrointestinal disorders) | 3 | 2
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 1
Accelerated hypertension (Vascular disorders) | 1 | 3
Accidental death (General disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 2 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Agitation (Psychiatric disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 2 | 0
Anal abscess (Infections and infestations) | 2 | 3
Anal fistula (Gastrointestinal disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Articular calcification (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthenia (General disorders) | 12 | 8
Atrioventricular block second degree (Cardiac disorders) | 2 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 1
Bronchitis (Infections and infestations) | 38 | 34
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 1
Bursitis infective (Infections and infestations) | 0 | 3
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Candida sepsis (Infections and infestations) | 1 | 0
Cardiac arrest (Cardiac disorders) | 27 | 28
Cardiac enzymes increased (Investigations) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 25 | 20
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 3 | 2
Cerebral haemorrhage traumatic (Injury, poisoning and procedural complications) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Chemical poisoning (Injury, poisoning and procedural complications) | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 1 | 0
Chordae tendinae rupture (Cardiac disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Completed suicide (Psychiatric disorders) | 2 | 1
Convulsion (Nervous system disorders) | 8 | 6
Cor pulmonale acute (Cardiac disorders) | 2 | 2
Coronary artery insufficiency (Cardiac disorders) | 2 | 2
Coronary artery occlusion (Cardiac disorders) | 2 | 2
Coronary artery stenosis (Cardiac disorders) | 4 | 6
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0
Cyst rupture (General disorders) | 0 | 1
Cystic lymphangioma (Congenital, familial and genetic disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Device capturing issue (General disorders) | 0 | 1
Device stimulation issue (General disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 2 | 4
Drug dispensing error (Injury, poisoning and procedural complications) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 31
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Electrocardiogram abnormal (Investigations) | 0 | 1
Embolic stroke (Nervous system disorders) | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 34
Exercise tolerance decreased (General disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 47 | 48
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Hantaviral infection (Infections and infestations) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 2
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7
Hepatitis A (Infections and infestations) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 3 | 4
Hypertensive heart disease (Cardiac disorders) | 2 | 2
Hypotension (Vascular disorders) | 20 | 12
Ileitis (Gastrointestinal disorders) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 5 | 2
Inflammation (General disorders) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 2
Jaundice (Hepatobiliary disorders) | 3 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lethargy (Nervous system disorders) | 1 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 2 | 2
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 8
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Malabsorption (Gastrointestinal disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 11 | 9
Meningitis (Infections and infestations) | 0 | 1
Meningorrhagia (Nervous system disorders) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 3 | 3
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 3 | 9
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Nail infection (Infections and infestations) | 0 | 1
Nail injury (Injury, poisoning and procedural complications) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Palpitations (Cardiac disorders) | 12 | 6
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 9
Parkinson's disease (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 5 | 0
Perineal infection (Infections and infestations) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 7 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 | 12
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 12 | 5
Pulmonary renal syndrome (Renal and urinary disorders) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelocystitis (Infections and infestations) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 3
Rectal abscess (Infections and infestations) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 | 18
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 6 | 9
Shock haemorrhagic (Vascular disorders) | 0 | 2
Sinus arrhythmia (Cardiac disorders) | 4 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 | 4
Spinal cord compression (Nervous system disorders) | 0 | 1
Subclavian artery aneurysm (Vascular disorders) | 0 | 1
Subdural effusion (Nervous system disorders) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 7
Tachyarrhythmia (Cardiac disorders) | 8 | 6
Tachycardia (Cardiac disorders) | 6 | 3
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Toothache (Gastrointestinal disorders) | 1 | 2
Trichiasis (Eye disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 2 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Viraemia (Infections and infestations) | 1 | 0
Vocal cord atrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin (N=9088) | Apixaban (N=9052)
Contusion (Injury, poisoning and procedural complications) | 299 | 479
Diarrhoea (Gastrointestinal disorders) | 580 | 581
Back pain (Musculoskeletal and connective tissue disorders) | 428 | 502
Cough (Respiratory, thoracic and mediastinal disorders) | 493 | 505
Headache (Nervous system disorders) | 480 | 485
Oedema peripheral (General disorders) | 607 | 661
Dizziness (Nervous system disorders) | 654 | 702
Urinary tract infection (Infections and infestations) | 471 | 501
Nasopharyngitis (Infections and infestations) | 763 | 779
Arthralgia (Musculoskeletal and connective tissue disorders) | 444 | 462
Bronchitis (Infections and infestations) | 473 | 493
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 583 | 633
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 547 | 666

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.